CLINICAL TRIAL: NCT02799472
Title: A Phase IIa, Double-Blind, Mechanistic Study of GSK3196165 in Combination With Methotrexate Therapy in Subjects With Active Rheumatoid Arthritis Despite Treatment With DMARDs
Brief Title: Mechanistic Study of GSK3196165 Plus Methotrexate (MTX) in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205180; 2015-004386-91 (EudraCT Number)
Record Dates: First submitted 2016-05-26; First posted 2016-06-14 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: GSK3196165; magnetic resonance imaging (MRI); disease-modifying antirheumatic drugs (DMARDs); granulocyte-macrophage colony stimulating factor (GM-CSF); Rheumatoid Arthritis; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab; Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK3196165 + MTX arm (Experimental): Subjects will receive GSK3196165 (initially weekly, then every other week) in combination with MTX (15-25 mg/week) and folic (or folinic) acid (>=5 mg/week).
  Interventions: Drug: GSK3196165; Drug: MTX; Drug: Folic (or folinic) acid
- Placebo + MTX arm (Placebo Comparator): Subjects will receive placebo (initially weekly, then every other week) in combination with MTX (15-25 mg/week) and folic (or folinic) acid (>=5 mg/week).
  Interventions: Drug: Placebo; Drug: MTX; Drug: Folic (or folinic) acid

INTERVENTIONS:
Drug: GSK3196165 — GSK3196165 is supplied as liquid and will be administered as SC injection.
  Arms: GSK3196165 + MTX arm
Drug: Placebo — 0.9% weight by volume (w/v) sodium chloride solution administered as SC injection.
  Arms: Placebo + MTX arm
Drug: MTX — Capsule, tablet or liquid administered orally or as SC injection.
Drug: Folic (or folinic) acid — Capsule, tablet or liquid and will be administered orally.

SUMMARY:
This study is designed to explore the activity of granulocyte-macrophage colony stimulating factor (GM-CSF) signaling pathway in subjects with rheumatoid arthritis (RA), the potential impact of inhibition of this axis by GSK3196165, and to evaluate whether there are any differences in the GM-CSF axis between subjects with early RA compared with those with more established disease. This study also aims to establish the potential impact of GSK3196165 on inflammatory structural joint damage in the hand/wrist using magnetic resonance imaging (MRI). This is a randomized Phase IIa, multi-center, double-blind, placebo-controlled parallel group study. Approximately 40 subjects with active RA despite treatment with disease-modifying antirheumatic drugs (DMARDs) (including conventional or biologic) will be randomized into the study, following a screening period of up to 6 weeks. The total treatment period is up to 10 weeks, with a 12-week follow-up period after the last dose (Week 22).

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years at the time of signing informed consent.
* Meets American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2010 RA Classification Criteria AND subject not diagnosed before age of 16 years.
* Functional class I, II or III defined by the 1992 ACR Classification of Functional Status in RA.
* Active disease as defined by:

  * Swollen joint count of >=4 (66-joint count) and tender joint count of >=4 (68-joint count) at screening and Day 1.

AND • Disease activity score for 28 different joints with C-reactive protein (CRP) value (DAS28[CRP]) >=3.2 at screening.

AND

• CRP >=3.0 milligrams (mg)/liter (L).

* Signs of inflammation such as synovitis in the MRI scan of the most-affected hand.
* Must be currently taking MTX (15-25 mg weekly) (oral/injected) for at least 12 weeks before screening, with no change in route of administration, with a stable and tolerated dose for >=4 weeks prior to Day 1. A stable dose of MTX >=7.5 mg/week is acceptable, if the MTX dose has been reduced for reasons of documented intolerance to MTX, example (e.g.) hepatic or hematologic toxicity, or per local requirement.
* Body weight >=45 kilograms (kg).
* Male or female subjects are eligible to participate so long as they meet and agree to abide by the contraceptive criteria.
* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.
* Willing to continue or initiate treatment with oral folic acid (at least 5 mg/week) or equivalent and be treated during the entire study (mandatory co-medication for MTX treatment).
* Diffusing capacity of the lung for carbon monoxide (DLCO) >=60% predicted; forced expiratory volume in 1 second (FEV1) >=70% predicted.
* No evidence of active or latent infection with Mycobacterium tuberculosis (TB).

Exclusion Criteria:

* Pregnant or lactating, or women planning to become pregnant or initiating breastfeeding.
* History of other inflammatory rheumatologic or autoimmune disorders, other than Sjögren's syndrome secondary to RA.
* History of any respiratory disease which (in the opinion of the investigator) would compromise subject safety or the ability of the subject to complete the study (e.g. significant interstitial lung disease, such as pulmonary fibrosis, chronic obstructive pulmonary disease (COPD), moderate-severe asthma, bronchiectasis, previous pulmonary alveolar proteinosis [PAP]).
* Clinically-significant (in the opinion of the investigator) persistent cough or clinically significant or unstable dyspnea that is unexplained.
* Significant unstable or uncontrolled acute or chronic disease which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* A history of malignancy.
* Contraindication to MRI scanning.
* Current/previous Hepatitis B virus (HBV), Hepatitis C virus (HCV) or human immunodeficiency virus (HIV) 1 or 2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (8):
  - GSK Investigational Site, El Cajon, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Houston, Texas
- Germany (2):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Püttlingen
- Poland (5):
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Nowa Sól
  - GSK Investigational Site, Piaseczno
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20745

REFERENCES:
- [Background] Genovese MC, Berkowitz M, Conaghan PG, Peterfy C, Davy K, Fisheleva E, Gupta A, Inman D, Janiczek R, Layton M, Mitchell N, Patel J, Roberts A, Saurigny D, Smith JE, Williamson R, Tak PP. MRI of the joint and evaluation of the granulocyte-macrophage colony-stimulating factor-CCL17 axis in patients with rheumatoid arthritis receiving otilimab: a phase 2a randomised mechanistic study. Lancet Rheumatol. 2020 Nov;2(11):e666-e676. doi: 10.1016/S2665-9913(20)30224-1. Epub 2020 Oct 7. PMID 38279363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 39 participants with active early/established Rheumatoid arthritis were randomized across 9 centers in 3 countries from 15 June 2016 to 30 October 2017.
Pre-assignment Details: Out of the 88 participants screened for this study, 49 participants were screen failures and 39 participants were randomized and received treatment in the study.
Groups:
- Placebo: Eligible participants received matching placebo subcutaneously (SC) into thigh or abdomen once weekly for 5 weeks, and then every other week until Week 10. In addition to placebo, participants also received methotrexate (MTX) 7.5-25 mg/week and folic (or folinic) acid >=5 mg/week during the combination treatment period.
- GSK3196165 180 mg: Eligible participants received GSK3196165 180 milligrams (mg) SC into thigh or abdomen once weekly for 5 weeks, and then every other week until Week 10. In addition to GSK3196165, participants also received MTX 7.5-5 mg/week and folic (or folinic) acid >=5 mg/week during the combination treatment period.
Period: Overall Study
Arm/Group | Placebo | GSK3196165 180 mg
Started | 11 | 28
Completed | 7 | 23
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants received matching placebo SC into thigh or abdomen once weekly for 5 weeks, and then every other week until Week 10. In addition to placebo, participants also received MTX 7.5-25 mg/week and folic (or folinic) acid >=5 mg/week during the combination treatment period.
- GSK3196165 180 mg: Eligible participants received GSK3196165 180 mg SC into thigh or abdomen once weekly for 5 weeks, and then every other week until Week 10. In addition to GSK3196165, participants also received MTX 7.5-5 mg/week and folic (or folinic) acid >=5 mg/week during the combination treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3196165 180 mg | Total
Number analyzed (Participants) | 11 | 28 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (11.57) | 59.1 (9.47) | 56.6 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 24 | 34
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 4 | 6
  White | 9 | 24 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Target Engagement Biomarkers- Soluble Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) Complexed to GSK3196165
Description: Blood samples were collected for markers which may influence rheumatoid arthritis. Target engagement biomarkers included soluble GM-CSF complexed to GSK3196165. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for GM-CSF - Complex log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Analysis was performed on Intent-to-Treat (ITT) Population which consisted of all participants who were randomized to treatment and who received at least one dose of study treatment. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week follow-up (FU) (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of GM-CSF complex
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of GM-CSF complex
  GM-CSF - Complex, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  GM-CSF - Complex, Week 1, n=9, 27 | 0.972 (35.98) | 13.799 (20.65)
  GM-CSF - Complex, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  GM-CSF - Complex, Week 2, n=8, 26 | 0.960 (31.23) | 31.056 (17.58)
  GM-CSF - Complex, Week 4, n=8, 27: number analyzed (Participants) | 8 | 27
  GM-CSF - Complex, Week 4, n=8, 27 | 0.959 (34.51) | 53.496 (18.55)
  GM-CSF - Complex, Week 6, n=7, 26: number analyzed (Participants) | 7 | 26
  GM-CSF - Complex, Week 6, n=7, 26 | 0.964 (40.96) | 46.620 (22.37)
  GM-CSF - Complex, Week 8, n=7, 24: number analyzed (Participants) | 7 | 24
  GM-CSF - Complex, Week 8, n=7, 24 | 0.964 (41.80) | 33.404 (22.47)
  GM-CSF - Complex, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  GM-CSF - Complex, Week 12, n=7, 24 | 0.970 (44.95) | 22.556 (24.38)
  GM-CSF - Complex, 12-Week FU, n=8, 21: number analyzed (Participants) | 8 | 21
  GM-CSF - Complex, 12-Week FU, n=8, 21 | 0.954 (20.80) | 1.176 (12.88)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; GM-CSF - Complex, Week 1; Test type: Other; p < 0.001, Repeated measures analysis; Ratio = 14.201, 95% CI 2-sided [6.251 to 32.262]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; GM-CSF - Complex, Week 2; Test type: Other; p < 0.001, Repeated measures analysis; Ratio = 32.360, 95% CI 2-sided [15.828 to 66.156]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; GM-CSF - Complex, Week 4; Test type: Other; p < 0.001, Repeated measures analysis; Ratio = 55.772, 95% CI 2-sided [25.646 to 121.287]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; GM-CSF - Complex, Week 6; Test type: Other; p < 0.001, Repeated measures analysis; Ratio = 48.336, 95% CI 2-sided [19.341 to 120.798]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; GM-CSF - Complex, Week 8; Test type: Other; p < 0.001, Repeated measures analysis; Ratio = 34.635, 95% CI 2-sided [13.690 to 87.629]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; GM-CSF - Complex, Week 12; Test type: Other; p < 0.001, Repeated measures analysis; Ratio = 23.249, 95% CI 2-sided [8.579 to 63.005]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; GM-CSF - Complex, 12-Week FU; Test type: Other; p = 0.401, Repeated measures analysis; Ratio = 1.233, 95% CI 2-sided [0.742 to 2.048]

2. Primary Outcome: Change From Baseline in Predictive Biomarkers: 14-3-3 ETA Protein, S100 Calcium Binding Protein (CBP) A8 and A9
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Predictive biomarkers included analysis of 14-3-3 ETA Protein, S100 CBP A8 and A9. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for 14-3-3 ETA Protein (mg/L) and S100 CBP A8 and A9 log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of predictive biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of predictive biomarker
  14-3-3 ETA Protein, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  14-3-3 ETA Protein, Week 1, n=9, 27 | 1.046 (3.88) | 0.986 (2.16)
  14-3-3 ETA Protein, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  14-3-3 ETA Protein, Week 2, n=8, 26 | 0.959 (12.14) | 0.986 (6.70)
  14-3-3 ETA Protein, Week 4, n=9, 26: number analyzed (Participants) | 9 | 26
  14-3-3 ETA Protein, Week 4, n=9, 26 | 1.128 (16.59) | 0.838 (9.55)
  14-3-3 ETA Protein, Week 6, n=7, 26: number analyzed (Participants) | 7 | 26
  14-3-3 ETA Protein, Week 6, n=7, 26 | 1.093 (15.55) | 0.833 (8.88)
  14-3-3 ETA Protein, Week 8, n=7, 23: number analyzed (Participants) | 7 | 23
  14-3-3 ETA Protein, Week 8, n=7, 23 | 0.950 (15.19) | 0.842 (8.48)
  14-3-3 ETA Protein, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  14-3-3 ETA Protein, Week 12, n=7, 24 | 1.131 (20.90) | 0.897 (11.89)
  14-3-3 ETA Protein, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  14-3-3 ETA Protein, 12-Week FU, n=7, 21 | 1.040 (24.06) | 0.893 (13.45)
  S100 CBP A8 and A9, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  S100 CBP A8 and A9, Week 1, n=9, 27 | 0.940 (15.20) | 0.939 (8.92)
  S100 CBP A8 and A9, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  S100 CBP A8 and A9, Week 2, n=8, 26 | 0.871 (15.28) | 0.823 (8.65)
  S100 CBP A8 and A9, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  S100 CBP A8 and A9, Week 4, n=9, 27 | 0.874 (19.20) | 0.889 (11.26)
  S100 CBP A8 and A9, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  S100 CBP A8 and A9, Week 6, n=7, 27 | 0.828 (21.92) | 0.812 (11.81)
  S100 CBP A8 and A9, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  S100 CBP A8 and A9, Week 8, n=7, 25 | 0.804 (21.04) | 0.857 (11.46)
  S100 CBP A8 and A9, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  S100 CBP A8 and A9, Week 12, n=7, 24 | 0.694 (21.61) | 0.879 (12.05)
  S100 CBP A8 and A9, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  S100 CBP A8 and A9, 12-Week FU, n=7, 21 | 0.582 (20.60) | 1.018 (11.83)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; 14-3-3 ETA Protein, Week 1; Test type: Other; p = 0.193, Repeated measures analysis; Ratio = 0.943, 95% CI 2-sided [0.861 to 1.032]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; 14-3-3 ETA Protein, Week 2; Test type: Other; p = 0.842, Repeated measures analysis; Ratio = 1.028, 95% CI 2-sided [0.776 to 1.362]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; 14-3-3 ETA Protein, Week 4; Test type: Other; p = 0.127, Repeated measures analysis; Ratio = 0.743, 95% CI 2-sided [0.505 to 1.093]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; 14-3-3 ETA Protein, Week 6; Test type: Other; p = 0.137, Repeated measures analysis; Ratio = 0.762, 95% CI 2-sided [0.531 to 1.095]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; 14-3-3 ETA Protein, Week 8; Test type: Other; p = 0.488, Repeated measures analysis; Ratio = 0.886, 95% CI 2-sided [0.623 to 1.259]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; 14-3-3 ETA Protein, Week 12; Test type: Other; p = 0.338, Repeated measures analysis; Ratio = 0.793, 95% CI 2-sided [0.488 to 1.290]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; 14-3-3 ETA Protein, 12-Week FU; Test type: Other; p = 0.582, Repeated measures analysis; Ratio = 0.859, 95% CI 2-sided [0.491 to 1.502]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; S100 CBP A8 and A9, Week 1; Test type: Other; p = 0.996, Repeated measures analysis; Ratio = 0.999, 95% CI 2-sided [0.699 to 1.427]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; S100 CBP A8 and A9, Week 2; Test type: Other; p = 0.745, Repeated measures analysis; Ratio = 0.944, 95% CI 2-sided [0.662 to 1.346]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; S100 CBP A8 and A9, Week 4; Test type: Other; p = 0.939, Repeated measures analysis; Ratio = 1.017, 95% CI 2-sided [0.649 to 1.593]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; S100 CBP A8 and A9, Week 6; Test type: Other; p = 0.937, Repeated measures analysis; Ratio = 0.981, 95% CI 2-sided [0.595 to 1.617]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; S100 CBP A8 and A9, Week 8; Test type: Other; p = 0.787, Repeated measures analysis; Ratio = 1.067, 95% CI 2-sided [0.659 to 1.727]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; S100 CBP A8 and A9, Week 12; Test type: Other; p = 0.342, Repeated measures analysis; Ratio = 1.267, 95% CI 2-sided [0.769 to 2.086]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; S100 CBP A8 and A9, 12-Week FU; Test type: Other; p = 0.026, Repeated measures analysis; Ratio = 1.748, 95% CI 2-sided [1.076 to 2.838]

3. Primary Outcome: Change From Baseline in Predictive Biomarkers: Amyloid A
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Predictive biomarkers included analysis of Amyloid A. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for Amyloid A log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Data has been presented for only those time points at which the samples were collected.
Time Frame: Baseline and Week 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of predictive biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of predictive biomarker
  Amyloid A, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Amyloid A, Week 12, n=7, 24 | 0.845 (49.31) | 0.653 (25.45)
  Amyloid A, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Amyloid A, 12-Week FU, n=7, 21 | 0.529 (35.12) | 0.623 (19.68)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Amyloid A, Week 12; Test type: Other; p = 0.632, Repeated measures analysis; Ratio = 0.774, 95% CI 2-sided [0.261 to 2.290]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Amyloid A, 12-Week FU; Test type: Other; p = 0.685, Repeated measures analysis; Ratio = 1.176, 95% CI 2-sided [0.519 to 2.663]

4. Primary Outcome: Change From Baseline in Predictive Biomarkers: Amyloid A, Chemokine (C-C Motif) Ligand 17, Chemokine (C-X-C Motif) Ligand 13, Interleukin 6, Macrophage-Derived Chemokine
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Predictive biomarkers included analysis of Chemokine (C-C Motif) Ligand 17 (CL17), Chemokine (C-X-C Motif) Ligand 13 (CL13), Interleukin 6, Macrophage-Derived Chemokine (MDC). Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for CL17, CL13, Interleukin 6, MDC log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Data has been presented for only those time points at which the samples were collected.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of predictive biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of predictive biomarker
  CL17, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  CL17, Week 1, n=9, 27 | 1.117 (18.81) | 0.773 (10.94)
  CL17, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  CL17, Week 2, n=8, 26 | 0.912 (24.37) | 0.651 (13.60)
  CL17, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  CL17, Week 4, n=9, 27 | 1.117 (21.91) | 0.679 (12.51)
  CL17, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  CL17, Week 6, n=7, 27 | 1.032 (24.38) | 0.779 (12.48)
  CL17, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  CL17, Week 8, n=7, 25 | 1.211 (20.63) | 0.675 (11.21)
  CL17, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  CL17, Week 12, n=7, 24 | 1.711 (24.96) | 0.890 (13.90)
  CL17, 12-Week FU, n=7, 20: number analyzed (Participants) | 7 | 20
  CL17, 12-Week FU, n=7, 20 | 1.434 (23.26) | 1.357 (13.59)
  CL13, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  CL13, Week 1, n=9, 27 | 1.198 (15.63) | 0.915 (8.87)
  CL13, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  CL13, Week 2, n=8, 26 | 1.090 (13.98) | 1.095 (7.78)
  CL13, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  CL13, Week 4, n=9, 27 | 0.947 (15.58) | 1.170 (8.90)
  CL13, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  CL13, Week 6, n=7, 27 | 0.839 (17.20) | 1.038 (8.91)
  CL13, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  CL13, Week 8, n=7, 25 | 0.913 (23.70) | 1.021 (12.38)
  CL13, Week 12, n=7,24: number analyzed (Participants) | 7 | 24
  CL13, Week 12, n=7,24 | 0.924 (31.17) | 1.077 (16.31)
  CL13, 12-Week FU, n=7,21: number analyzed (Participants) | 7 | 21
  CL13, 12-Week FU, n=7,21 | 0.774 (27.82) | 1.224 (15.04)
  Interleukin 6, Week 1, n=9, 26: number analyzed (Participants) | 9 | 26
  Interleukin 6, Week 1, n=9, 26 | 1.179 (27.92) | 1.064 (16.38)
  Interleukin 6, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Interleukin 6, Week 2, n=8, 26 | 1.153 (29.33) | 0.830 (16.63)
  Interleukin 6, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Interleukin 6, Week 4, n=9, 27 | 0.986 (26.22) | 0.811 (15.10)
  Interleukin 6, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Interleukin 6, Week 6, n=7, 27 | 1.136 (24.95) | 0.748 (13.51)
  Interleukin 6, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Interleukin 6, Week 8, n=7, 25 | 1.275 (23.65) | 0.872 (13.35)
  Interleukin 6, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Interleukin 6, Week 12, n=7, 24 | 0.770 (21.89) | 0.939 (12.35)
  Interleukin 6, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Interleukin 6, 12-Week FU, n=7, 21 | 0.817 (33.13) | 1.308 (18.63)
  MDC, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  MDC, Week 1, n=9, 27 | 0.987 (5.02) | 0.914 (2.89)
  MDC, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  MDC, Week 2, n=8, 26 | 0.925 (7.33) | 0.911 (4.15)
  MDC, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  MDC, Week 4, n=9, 27 | 0.936 (8.13) | 0.895 (4.67)
  MDC, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  MDC, Week 6, n=7, 27 | 0.984 (8.38) | 0.994 (4.48)
  MDC, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  MDC, Week 8, n=7, 25 | 1.049 (9.36) | 0.899 (5.09)
  MDC, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  MDC, Week 12, n=7, 24 | 1.245 (9.51) | 1.058 (5.23)
  MDC, 12-Week FU, n=7, 20: number analyzed (Participants) | 7 | 20
  MDC, 12-Week FU, n=7, 20 | 1.303 (12.66) | 1.321 (7.53)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; CL17, Week 1; Test type: Other; p = 0.097, Repeated measures analysis; Ratio = 0.692, 95% CI 2-sided [0.445 to 1.074]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; CL17, Week 2; Test type: Other; p = 0.229, Repeated measures analysis; Ratio = 0.713, 95% CI 2-sided [0.407 to 1.249]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; CL17, Week 4; Test type: Other; p = 0.055, Repeated measures analysis; Ratio = 0.608, 95% CI 2-sided [0.365 to 1.012]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; CL17, Week 6; Test type: Other; p = 0.307, Repeated measures analysis; Ratio = 0.755, 95% CI 2-sided [0.435 to 1.309]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; CL17, Week 8; Test type: Other; p = 0.017, Repeated measures analysis; Ratio = 0.557, 95% CI 2-sided [0.348 to 0.894]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.026, Repeated measures analysis; Ratio = 0.520, 95% CI 2-sided [0.294 to 0.922]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; CL17, 12-Week FU; Test type: Other; p = 0.839, Repeated measures analysis; Ratio = 0.947, 95% CI 2-sided [0.548 to 1.636]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; CL13, Week 1; Test type: Other; p = 0.142, Repeated measures analysis; Ratio = 0.764, 95% CI 2-sided [0.530 to 1.100]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; CL13, Week 2; Test type: Other; p = 0.976, Repeated measures analysis; Ratio = 1.005, 95% CI 2-sided [0.726 to 1.390]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; CL13, Week 4; Test type: Other; p = 0.244, Repeated measures analysis; Ratio = 1.236, 95% CI 2-sided [0.859 to 1.778]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; CL13, Week 6; Test type: Other; p = 0.278, Repeated measures analysis; Ratio = 1.237, 95% CI 2-sided [0.836 to 1.830]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; CL13, Week 8; Test type: Other; p = 0.677, Repeated measures analysis; Ratio = 1.118, 95% CI 2-sided [0.651 to 1.920]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; CL13, Week 12; Test type: Other; p = 0.661, Repeated measures analysis; Ratio = 1.165, 95% CI 2-sided [0.573 to 2.369]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; CL13, 12-Week FU; Test type: Other; p = 0.154, Repeated measures analysis; Ratio = 1.581, 95% CI 2-sided [0.832 to 3.007]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; Interleukin 6, Week 1; Test type: Other; p = 0.751, Repeated measures analysis; Ratio = 0.903, 95% CI 2-sided [0.471 to 1.729]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 180 mg; Interleukin 6, Week 2; Test type: Other; p = 0.330, Repeated measures analysis; Ratio = 0.720, 95% CI 2-sided [0.367 to 1.413]
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 180 mg; Interleukin 6, Week 4; Test type: Other; p = 0.519, Repeated measures analysis; Ratio = 0.822, 95% CI 2-sided [0.447 to 1.512]
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 180 mg; Interleukin 6, Week 6; Test type: Other; p = 0.147, Repeated measures analysis; Ratio = 0.659, 95% CI 2-sided [0.372 to 1.167]
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 180 mg; Interleukin 6, Week 8; Test type: Other; p = 0.166, Repeated measures analysis; Ratio = 0.684, 95% CI 2-sided [0.396 to 1.180]
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 180 mg; Interleukin 6, Week 12; Test type: Other; p = 0.432, Repeated measures analysis; Ratio = 1.221, 95% CI 2-sided [0.734 to 2.031]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 180 mg; Interleukin 6, 12-Week FU; Test type: Other; p = 0.216, Repeated measures analysis; Ratio = 1.602, 95% CI 2-sided [0.750 to 3.423]
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 180 mg; MDC, Week 1; Test type: Other; p = 0.195, Repeated measures analysis; Ratio = 0.926, 95% CI 2-sided [0.823 to 1.042]
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 180 mg; MDC, Week 2; Test type: Other; p = 0.851, Repeated measures analysis; Ratio = 0.984, 95% CI 2-sided [0.829 to 1.168]
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 180 mg; MDC, Week 4; Test type: Other; p = 0.637, Repeated measures analysis; Ratio = 0.956, 95% CI 2-sided [0.790 to 1.158]
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 180 mg; MDC, Week 6; Test type: Other; p = 0.915, Repeated measures analysis; Ratio = 1.010, 95% CI 2-sided [0.833 to 1.225]
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 180 mg; MDC, Week 8; Test type: Other; p = 0.157, Repeated measures analysis; Ratio = 0.857, 95% CI 2-sided [0.690 to 1.064]
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 180 mg; MDC, Week 12; Test type: Other; p = 0.142, Repeated measures analysis; Ratio = 0.849, 95% CI 2-sided [0.681 to 1.059]
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 180 mg; MDC, 12-Week FU; Test type: Other; p = 0.929, Repeated measures analysis; Ratio = 1.013, 95% CI 2-sided [0.745 to 1.378]

5. Primary Outcome: Change From Baseline in Predictive Biomarkers: Chitinase 3 Like 1, Matrix Metalloproteinase 3 (MMP-3)
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Predictive biomarkers included analysis of Chitinase 3 Like 1 and MMP-3. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for Chitinase 3 Like 1 and MMP-3 log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of predictive biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of predictive biomarker
  Chitinase 3 Like 1, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  Chitinase 3 Like 1, Week 1, n=9, 27 | 1.033 (13.97) | 0.917 (8.13)
  Chitinase 3 Like 1, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Chitinase 3 Like 1, Week 2, n=8, 26 | 1.013 (15.05) | 0.966 (8.55)
  Chitinase 3 Like 1, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Chitinase 3 Like 1, Week 4, n=9, 27 | 0.961 (17.14) | 1.088 (9.96)
  Chitinase 3 Like 1, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Chitinase 3 Like 1, Week 6, n=7, 27 | 0.897 (17.08) | 1.031 (8.80)
  Chitinase 3 Like 1, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Chitinase 3 Like 1, Week 8, n=7, 25 | 0.851 (18.24) | 0.947 (9.70)
  Chitinase 3 Like 1, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Chitinase 3 Like 1, Week 12, n=7, 24 | 1.066 (21.53) | 1.071 (11.64)
  Chitinase 3 Like 1, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Chitinase 3 Like 1, 12-Week FU, n=7, 21 | 0.735 (16.87) | 1.019 (9.75)
  MMP 3, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  MMP 3, Week 1, n=9, 27 | 1.076 (6.72) | 0.984 (3.88)
  MMP-3, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  MMP-3, Week 2, n=8, 26 | 1.067 (7.26) | 1.024 (4.09)
  MMP-3, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  MMP-3, Week 4, n=9, 27 | 1.112 (8.30) | 1.016 (4.73)
  MMP-3, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  MMP-3, Week 6, n=7, 27 | 1.005 (26.26) | 0.804 (13.44)
  MMP-3, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  MMP-3, Week 8, n=7, 25 | 0.939 (15.43) | 1.088 (8.21)
  MMP-3, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  MMP-3, Week 12, n=7, 24 | 1.000 (13.57) | 0.951 (7.35)
  MMP-3, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  MMP-3, 12-Week FU, n=7, 21 | 0.803 (16.05) | 0.984 (9.00)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Chitinase 3 Like 1, Week 1; Test type: Other; p = 0.463, Repeated measures analysis; Ratio = 0.887, 95% CI 2-sided [0.640 to 1.231]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Chitinase 3 Like 1, Week 2; Test type: Other; p = 0.782, Repeated measures analysis; Ratio = 0.953, 95% CI 2-sided [0.672 to 1.352]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; Chitinase 3 Like 1, Week 4; Test type: Other; p = 0.533, Repeated measures analysis; Ratio = 1.132, 95% CI 2-sided [0.759 to 1.690]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; Chitinase 3 Like 1, Week 6; Test type: Other; p = 0.473, Repeated measures analysis; Ratio = 1.149, 95% CI 2-sided [0.779 to 1.694]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; Chitinase 3 Like 1, Week 8; Test type: Other; p = 0.608, Repeated measures analysis; Ratio = 1.112, 95% CI 2-sided [0.733 to 1.687]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; Chitinase 3 Like 1, Week 12; Test type: Other; p = 0.985, Repeated measures analysis; Ratio = 1.005, 95% CI 2-sided [0.613 to 1.645]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; Chitinase 3 Like 1, 12-Week FU; Test type: Other; p = 0.102, Repeated measures analysis; Ratio = 1.386, 95% CI 2-sided [0.934 to 2.057]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; MMP-3, Week 1; Test type: Other; p = 0.259, Repeated measures analysis; Ratio = 0.915, 95% CI 2-sided [0.781 to 1.071]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; MMP-3, Week 2; Test type: Other; p = 0.621, Repeated measures analysis; Ratio = 0.959, 95% CI 2-sided [0.809 to 1.137]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; MMP-3, Week 4; Test type: Other; p = 0.354, Repeated measures analysis; Ratio = 0.914, 95% CI 2-sided [0.752 to 1.110]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; MMP-3, Week 6; Test type: Other; p = 0.448, Repeated measures analysis; Ratio = 0.800, 95% CI 2-sided [0.443 to 1.444]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; MMP-3, Week 8; Test type: Other; p = 0.402, Repeated measures analysis; Ratio = 1.160, 95% CI 2-sided [0.813 to 1.653]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; MMP-3, Week 12; Test type: Other; p = 0.745, Repeated measures analysis; Ratio = 0.951, 95% CI 2-sided [0.695 to 1.301]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; MMP-3, 12-Week FU; Test type: Other; p = 0.279, Repeated measures analysis; Ratio = 1.226, 95% CI 2-sided [0.837 to 1.796]

6. Primary Outcome: Change From Baseline in Cartilage Biomarkers
Description: Blood samples were collected and analyzed for markers that may be predictive of rheumatoid arthritis disease activity. Cartilage biomarkers included analysis of ARGS Neo-Epitope, Citrullinated MMP-Degraded Vimentin (CMDV), MMP-Degraded C Reactive Protein (CRP), MMP-Degraded Type I Collagen (MD1C), MMP-Degraded Type II Collagen (MD2C), MMP-Degraded Type III Collagen (MD3C). Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for ARGS Neo-Epitope, Citrullinated MMP-Degraded Vimentin, MMP-Degraded CRP, MMP-Degraded Type I Collagen, MMP-Degraded Type II Collagen and MMP-Degraded Type III Collagen log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of cartilage biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of cartilage biomarker
  ARGS Neo-Epitope, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  ARGS Neo-Epitope, Week 1, n=9, 27 | 0.979 (16.10) | 1.075 (9.67)
  ARGS Neo-Epitope, Week 2, n=8, 25: number analyzed (Participants) | 8 | 25
  ARGS Neo-Epitope, Week 2, n=8, 25 | 0.790 (17.38) | 1.249 (9.87)
  ARGS Neo-Epitope, Week 4, n=8, 26: number analyzed (Participants) | 8 | 26
  ARGS Neo-Epitope, Week 4, n=8, 26 | 0.904 (17.02) | 1.104 (10.05)
  ARGS Neo-Epitope, Week 6, n=6, 26: number analyzed (Participants) | 6 | 26
  ARGS Neo-Epitope, Week 6, n=6, 26 | 0.894 (14.28) | 1.164 (7.82)
  ARGS Neo-Epitope, Week 8, n=7, 24: number analyzed (Participants) | 7 | 24
  ARGS Neo-Epitope, Week 8, n=7, 24 | 0.854 (26.42) | 1.238 (14.20)
  ARGS Neo-Epitope, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  ARGS Neo-Epitope, Week 12, n=7, 24 | 0.913 (13.97) | 1.156 (7.78)
  ARGS Neo-Epitope, 12-Week FU, n=8, 21: number analyzed (Participants) | 8 | 21
  ARGS Neo-Epitope, 12-Week FU, n=8, 21 | 1.129 (17.44) | 1.124 (9.86)
  CMDV, Week 1,n=9,27: number analyzed (Participants) | 9 | 27
  CMDV, Week 1,n=9,27 | 0.981 (24.12) | 0.876 (13.80)
  CMDV,Week 2,n=8,26: number analyzed (Participants) | 8 | 26
  CMDV,Week 2,n=8,26 | 0.820 (28.46) | 0.714 (15.89)
  CMDV, Week 4,n=9,27: number analyzed (Participants) | 9 | 27
  CMDV, Week 4,n=9,27 | 0.715 (27.30) | 0.801 (15.52)
  CMDV, Week 6,n=7,27: number analyzed (Participants) | 7 | 27
  CMDV, Week 6,n=7,27 | 1.099 (30.47) | 0.726 (15.94)
  CMDV, Week 8,n=7,25: number analyzed (Participants) | 7 | 25
  CMDV, Week 8,n=7,25 | 0.929 (24.72) | 0.759 (13.39)
  CMDV, Week12,n=7,24: number analyzed (Participants) | 7 | 24
  CMDV, Week12,n=7,24 | 1.123 (29.34) | 0.917 (16.00)
  CMDV, 12-Week FU,n=7,21: number analyzed (Participants) | 7 | 21
  CMDV, 12-Week FU,n=7,21 | 0.936 (28.05) | 0.769 (15.81)
  MMP-Degraded CRP, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  MMP-Degraded CRP, Week 1, n=9, 27 | 0.971 (6.83) | 1.021 (3.99)
  MMP-Degraded CRP, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  MMP-Degraded CRP, Week 2, n=8, 26 | 0.970 (5.55) | 1.000 (3.07)
  MMP-Degraded CRP, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  MMP-Degraded CRP, Week 4, n=9, 27 | 0.992 (6.01) | 1.004 (3.49)
  MMP-Degraded CRP, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  MMP-Degraded CRP, Week 6, n=7, 27 | 1.122 (6.55) | 1.099 (3.50)
  MMP-Degraded CRP, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  MMP-Degraded CRP, Week 8, n=7, 25 | 0.977 (7.37) | 1.087 (4.05)
  MMP-Degraded CRP, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  MMP-Degraded CRP, Week 12, n=7, 24 | 1.006 (7.13) | 1.108 (3.95)
  MMP-Degraded CRP, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  MMP-Degraded CRP, 12-Week FU, n=7, 21 | 1.075 (8.01) | 1.129 (4.48)
  MD1C, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  MD1C, Week 1, n=9, 27 | 1.079 (9.60) | 0.858 (5.63)
  MD1C, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  MD1C, Week 2, n=8, 26 | 1.028 (11.98) | 0.907 (6.63)
  MD1C, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  MD1C, Week 4, n=9, 27 | 1.142 (14.57) | 0.896 (8.35)
  MD1C, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  MD1C, Week 6, n=7, 27 | 1.392 (12.64) | 0.889 (6.98)
  MD1C, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  MD1C, Week 8, n=7, 25 | 1.131 (13.05) | 0.904 (7.23)
  MD1C, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  MD1C, Week 12, n=7, 24 | 1.148 (13.74) | 1.023 (7.81)
  MD1C, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  MD1C, 12-Week FU, n=7, 21 | 1.095 (14.21) | 0.952 (8.31)
  MD2C, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  MD2C, Week 1, n=9, 27 | 1.059 (11.83) | 1.038 (6.88)
  MD2C, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  MD2C, Week 2, n=8, 26 | 1.046 (11.27) | 1.015 (6.28)
  MD2C, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  MD2C, Week 4, n=9, 27 | 1.035 (10.18) | 1.003 (5.86)
  MD2C, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  MD2C, Week 6, n=7, 27 | 1.158 (12.07) | 1.064 (6.30)
  MD2C, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  MD2C, Week 8, n=7, 25 | 1.091 (11.42) | 1.023 (6.12)
  MD2C, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  MD2C, Week 12, n=7, 24 | 1.174 (10.73) | 1.072 (5.87)
  MD2C, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  MD2C, 12-Week FU, n=7, 21 | 1.338 (13.10) | 1.041 (7.50)
  MD3C, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  MD3C, Week 1, n=9, 27 | 0.950 (6.44) | 0.959 (3.74)
  MD3C, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  MD3C, Week 2, n=8, 26 | 0.920 (6.82) | 0.954 (3.91)
  MD3C, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  MD3C, Week 4, n=9, 27 | 0.940 (8.06) | 0.886 (4.68)
  MD3C, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  MD3C, Week 6, n=7, 27 | 1.013 (8.09) | 0.894 (4.34)
  MD3C, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  MD3C, Week 8, n=7, 25 | 0.918 (9.04) | 0.881 (4.84)
  MD3C, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  MD3C, Week 12, n=7, 24 | 0.929 (9.28) | 0.910 (5.08)
  MD3C, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  MD3C, 12-Week FU, n=7, 21 | 0.847 (9.75) | 0.910 (5.46)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; ARGS Neo-Epitope, Week 1; Test type: Other; p = 0.621, Repeated measures analysis; Ratio = 1.098, 95% CI 2-sided [0.750 to 1.606]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; ARGS Neo-Epitope, Week 2; Test type: Other; p = 0.031, Repeated measures analysis; Ratio = 1.581, 95% CI 2-sided [1.046 to 2.388]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; ARGS Neo-Epitope, Week 4; Test type: Other; p = 0.317, Repeated measures analysis; Ratio = 1.222, 95% CI 2-sided [0.817 to 1.827]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; ARGS Neo-Epitope, Week 6; Test type: Other; p = 0.113, Repeated measures analysis; Ratio = 1.302, 95% CI 2-sided [0.936 to 1.810]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; ARGS Neo-Epitope, Week 8; Test type: Other; p = 0.217, Repeated measures analysis; Ratio = 1.450, 95% CI 2-sided [0.795 to 2.645]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; ARGS Neo-Epitope, Week 12; Test type: Other; p = 0.147, Repeated measures analysis; Ratio = 1.266, 95% CI 2-sided [0.916 to 1.750]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; ARGS Neo-Epitope, 12-Week FU; Test type: Other; p = 0.985, Repeated measures analysis; Ratio = 0.996, 95% CI 2-sided [0.662 to 1.499]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; CMDV, Week 1; Test type: Other; p = 0.681, Repeated measures analysis; Ratio = 0.892, 95% CI 2-sided [0.511 to 1.560]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; CMDV, Week 2; Test type: Other; p = 0.668, Repeated measures analysis; Ratio = 0.870, 95% CI 2-sided [0.454 to 1.669]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; CMDV, Week 4; Test type: Other; p = 0.717, Repeated measures analysis; Ratio = 1.120, 95% CI 2-sided [0.597 to 2.101]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; CMDV, Week 6; Test type: Other; p = 0.227, Repeated measures analysis; Ratio = 0.661, 95% CI 2-sided [0.333 to 1.310]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; CMDV, Week 8; Test type: Other; p = 0.471, Repeated measures analysis; Ratio = 0.817, 95% CI 2-sided [0.464 to 1.437]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; CMDV, Week 12; Test type: Other; p = 0.541, Repeated measures analysis; Ratio = 0.816, 95% CI 2-sided [0.417 to 1.597]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; CMDV, 12-Week FU; Test type: Other; p = 0.544, Repeated measures analysis; Ratio = 0.822, 95% CI 2-sided [0.422 to 1.602]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; MMP-Degraded CRP, Week 1; Test type: Other; p = 0.537, Repeated measures analysis; Ratio = 1.051, 95% CI 2-sided [0.895 to 1.233]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 180 mg; MMP-Degraded CRP, Week 2; Test type: Other; p = 0.635, Repeated measures analysis; Ratio = 1.031, 95% CI 2-sided [0.906 to 1.173]
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 180 mg; MMP-Degraded CRP, Week 4; Test type: Other; p = 0.866, Repeated measures analysis; Ratio = 1.012, 95% CI 2-sided [0.879 to 1.165]
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 180 mg; MMP-Degraded CRP, Week 6; Test type: Other; p = 0.780, Repeated measures analysis; Ratio = 0.979, 95% CI 2-sided [0.842 to 1.139]
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 180 mg; MMP-Degraded CRP, Week 8; Test type: Other; p = 0.212, Repeated measures analysis; Ratio = 1.113, 95% CI 2-sided [0.938 to 1.320]
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 180 mg; MMP-Degraded CRP, Week 12; Test type: Other; p = 0.242, Repeated measures analysis; Ratio = 1.102, 95% CI 2-sided [0.934 to 1.300]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 180 mg; MMP-Degraded CRP, 12-Week FU; Test type: Other; p = 0.597, Repeated measures analysis; Ratio = 1.050, 95% CI 2-sided [0.870 to 1.267]
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 180 mg; MD1C, Week 1; Test type: Other; p = 0.047, Repeated measures analysis; Ratio = 0.795, 95% CI 2-sided [0.634 to 0.997]
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 180 mg; MD1C, Week 2; Test type: Other; p = 0.367, Repeated measures analysis; Ratio = 0.883, 95% CI 2-sided [0.668 to 1.165]
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 180 mg; MD1C, Week 4; Test type: Other; p = 0.155, Repeated measures analysis; Ratio = 0.784, 95% CI 2-sided [0.558 to 1.102]
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 180 mg; MD1C, Week 6; Test type: Other; p = 0.004, Repeated measures analysis; Ratio = 0.638, 95% CI 2-sided [0.477 to 0.855]
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 180 mg; MD1C, Week 8; Test type: Other; p = 0.140, Repeated measures analysis; Ratio = 0.799, 95% CI 2-sided [0.591 to 1.080]
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 180 mg; MD1C, Week 12; Test type: Other; p = 0.470, Repeated measures analysis; Ratio = 0.891, 95% CI 2-sided [0.647 to 1.228]
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 180 mg; MD1C, 12-Week FU; Test type: Other; p = 0.401, Repeated measures analysis; Ratio = 0.869, 95% CI 2-sided [0.621 to 1.217]
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 180 mg; MD2C, Week 1; Test type: Other; p = 0.887, Repeated measures analysis; Ratio = 0.981, 95% CI 2-sided [0.742 to 1.296]
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 180 mg; MD2C, Week 2; Test type: Other; p = 0.814, Repeated measures analysis; Ratio = 0.970, 95% CI 2-sided [0.744 to 1.263]
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; MD2C, Week 4; Test type: Other; p = 0.794, Repeated measures analysis; Ratio = 0.969, 95% CI 2-sided [0.762 to 1.233]
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 180 mg; MD2C, Week 6; Test type: Other; p = 0.539, Repeated measures analysis; Ratio = 0.919, 95% CI 2-sided [0.696 to 1.213]
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 180 mg; MD2C, Week 8; Test type: Other; p = 0.623, Repeated measures analysis; Ratio = 0.937, 95% CI 2-sided [0.719 to 1.221]
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 180 mg; MD2C, Week 12; Test type: Other; p = 0.467, Repeated measures analysis; Ratio = 0.913, 95% CI 2-sided [0.711 to 1.173]
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; MD2C, 12-Week FU; Test type: Other; p = 0.108, Repeated measures analysis; Ratio = 0.778, 95% CI 2-sided [0.570 to 1.061]
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 180 mg; MD3C, Week 1; Test type: Other; p = 0.897, Repeated measures analysis; Ratio = 1.010, 95% CI 2-sided [0.868 to 1.175]
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; MD3C, Week 2; Test type: Other; p = 0.644, Repeated measures analysis; Ratio = 1.037, 95% CI 2-sided [0.884 to 1.218]
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 180 mg; MD3C, Week 4; Test type: Other; p = 0.530, Repeated measures analysis; Ratio = 0.943, 95% CI 2-sided [0.780 to 1.139]
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; MD3C, Week 6; Test type: Other; p = 0.182, Repeated measures analysis; Ratio = 0.882, 95% CI 2-sided [0.733 to 1.063]
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 180 mg; MD3C, Week 8; Test type: Other; p = 0.691, Repeated measures analysis; Ratio = 0.960, 10% CI 2-sided [0.779 to 1.182]
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; MD3C, Week 12; Test type: Other; p = 0.843, Repeated measures analysis; Ratio = 0.979, 95% CI 2-sided [0.790 to 1.214]
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 180 mg; MD3C, 12-Week FU; Test type: Other; p = 0.524, Repeated measures analysis; Ratio = 1.075, 95% CI 2-sided [0.855 to 1.351]

7. Primary Outcome: Change From Baseline in Flow Cytometry: Helper/Suppressor Cells
Description: Whole blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Flow cytometry assessment included assessment of Helper/Suppressor. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for Helper/Suppressor log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of Helper/Suppressor cells
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of Helper/Suppressor cells
  Helper/Suppressor, Week 1, n=8, 25: number analyzed (Participants) | 8 | 25
  Helper/Suppressor, Week 1, n=8, 25 | 1.024 (6.98) | 0.976 (4.00)
  Helper/Suppressor, Week 4, n=8, 25: number analyzed (Participants) | 8 | 25
  Helper/Suppressor, Week 4, n=8, 25 | 1.053 (7.18) | 0.998 (4.11)
  Helper/Suppressor, Week 12, n=6, 25: number analyzed (Participants) | 6 | 25
  Helper/Suppressor, Week 12, n=6, 25 | 1.040 (6.83) | 1.088 (3.49)
  Helper/Suppressor, 12-Week FU, n=6, 21: number analyzed (Participants) | 6 | 21
  Helper/Suppressor, 12-Week FU, n=6, 21 | 1.051 (8.99) | 1.065 (4.88)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Helper/Suppressor, Week 1; Test type: Other; p = 0.558, Repeated measures analysis; Ratio = 0.953, 95% CI 2-sided [0.809 to 1.123]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Helper/Suppressor, Week 4; Test type: Other; p = 0.515, Repeated measures analysis; Ratio = 0.947, 95% CI 2-sided [0.801 to 1.120]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; Helper/Suppressor, Week 12; Test type: Other; p = 0.565, Repeated measures analysis; Ratio = 1.046, 95% CI 2-sided [0.895 to 1.222]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; Helper/Suppressor, 12-Week FU; Test type: Other; p = 0.897, Repeated measures analysis; Ratio = 1.013, 95% CI 2-sided [0.822 to 1.249]

8. Primary Outcome: Change From Baseline in Flow Cytometry: 6 Colour TB Natural Killer (NK) Panel- CD16+CD56+, CD19, CD3, CD3+CD4+
Description: Whole blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Flow cytometry assessment included assessment of cluster of differentiation (CD)16+CD56+, CD19, CD3, CD3+CD4+. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Repeated measures analysis adjusted for CD16+CD56+, CD19, CD3, CD3+CD4+, CD3+CD8+ and T Cell B Cell NKL log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of biomarker
  CD16+CD56+, Week 1, n=8, 25: number analyzed (Participants) | 8 | 25
  CD16+CD56+, Week 1, n=8, 25 | 0.989 (11.39) | 1.025 (6.30)
  CD16+CD56+, Week 4, n=8, 25: number analyzed (Participants) | 8 | 25
  CD16+CD56+, Week 4, n=8, 25 | 1.163 (12.97) | 0.951 (7.25)
  CD16+CD56+, Week 12, n=6, 25: number analyzed (Participants) | 6 | 25
  CD16+CD56+, Week 12, n=6, 25 | 1.193 (15.49) | 0.911 (7.81)
  CD16+CD56+, 12-Week FU, n=6, 21: number analyzed (Participants) | 6 | 21
  CD16+CD56+, 12-Week FU, n=6, 21 | 1.298 (15.10) | 0.920 (7.98)
  CD19, Week 1, n=8, 25: number analyzed (Participants) | 8 | 25
  CD19, Week 1, n=8, 25 | 0.880 (11.05) | 0.984 (6.23)
  CD19, Week 4, n=8, 25: number analyzed (Participants) | 8 | 25
  CD19, Week 4, n=8, 25 | 1.090 (15.31) | 0.971 (8.60)
  CD19, Week 12, n=6, 25: number analyzed (Participants) | 6 | 25
  CD19, Week 12, n=6, 25 | 1.054 (12.26) | 1.003 (6.51)
  CD19, Week 22, n=6, 21: number analyzed (Participants) | 6 | 21
  CD19, Week 22, n=6, 21 | 0.980 (17.75) | 0.938 (9.75)
  CD3, Week 1, n=8, 25: number analyzed (Participants) | 8 | 25
  CD3, Week 1, n=8, 25 | 0.918 (8.73) | 0.994 (4.95)
  CD3, Week 4, n=8, 25: number analyzed (Participants) | 8 | 25
  CD3, Week 4, n=8, 25 | 0.997 (11.79) | 0.934 (6.66)
  CD3, Week 12, n=6, 25: number analyzed (Participants) | 6 | 25
  CD3, Week 12, n=6, 25 | 0.912 (9.01) | 0.992 (4.60)
  CD3, 12-Week FU, n=6, 21: number analyzed (Participants) | 6 | 21
  CD3, 12-Week FU, n=6, 21 | 0.931 (9.17) | 0.989 (4.98)
  CD3+CD4+, Week 1, n=8, 25: number analyzed (Participants) | 8 | 25
  CD3+CD4+, Week 1, n=8, 25 | 0.926 (9.56) | 0.991 (5.42)
  CD3+CD4+, Week 4, n=8, 25: number analyzed (Participants) | 8 | 25
  CD3+CD4+, Week 4, n=8, 25 | 1.028 (12.80) | 0.933 (7.23)
  CD3+CD4+, Week 12, n=6, 25: number analyzed (Participants) | 6 | 25
  CD3+CD4+, Week 12, n=6, 25 | 0.952 (9.69) | 1.013 (4.94)
  CD3+CD4+, 12-Week FU, n=6, 21: number analyzed (Participants) | 6 | 21
  CD3+CD4+, 12-Week FU, n=6, 21 | 0.970 (9.92) | 1.000 (5.37)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; CD16+CD56+, Week 1; Test type: Other; p = 0.786, Repeated measures analysis; Ratio = 1.037, 95% CI 2-sided [0.794 to 1.354]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; CD16+CD56+, Week 4; Test type: Other; p = 0.188, Repeated measures analysis; Ratio = 0.818, 95% CI 2-sided [0.603 to 1.109]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; CD16+CD56+, Week 12; Test type: Other; p = 0.129, Repeated measures analysis; Ratio = 0.763, 95% CI 2-sided [0.536 to 1.087]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; CD16+CD56+, 12-Week FU; Test type: Other; p = 0.054, Repeated measures analysis; Ratio = 0.709, 95% CI 2-sided [0.499 to 1.006]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; CD19, Week 1; Test type: Other; p = 0.383, Repeated measures analysis; Ratio = 1.119, 95% CI 2-sided [0.863 to 1.450]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; CD19, Week 4; Test type: Other; p = 0.510, Repeated measures analysis; Ratio = 0.890, 95% CI 2-sided [0.623 to 1.271]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; CD19, Week 12; Test type: Other; p = 0.724, Repeated measures analysis; Ratio = 0.952, 95% CI 2-sided [0.718 to 1.262]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; CD19, 12-Week FU; Test type: Other; p = 0.831, Repeated measures analysis; Ratio = 0.958, 95% CI 2-sided [0.635 to 1.443]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; CD3, Week 1; Test type: Other; p = 0.437, Repeated measures analysis; Ratio = 1.082, 95% CI 2-sided [0.882 to 1.328]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; CD3, Week 4; Test type: Other; p = 0.632, Repeated measures analysis; Ratio = 0.937, 95% CI 2-sided [0.711 to 1.234]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; CD3, Week 12; Test type: Other; p = 0.413, Repeated measures analysis; Ratio = 1.088, 95% CI 2-sided [0.885 to 1.336]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; CD3, 12-Week FU; Test type: Other; p = 0.567, Repeated measures analysis; Ratio = 1.062, 95% CI 2-sided [0.858 to 1.316]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+, Week 1; Test type: Other; p = 0.547, Repeated measures analysis; Ratio = 1.069, 95% CI 2-sided [0.855 to 1.338]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+, Week 4; Test type: Other; p = 0.512, Repeated measures analysis; Ratio = 0.907, 95% CI 2-sided [0.673 to 1.223]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+, Week 12; Test type: Other; p = 0.573, Repeated measures analysis; Ratio = 1.064, 95% CI 2-sided [0.853 to 1.328]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+, 12-Week FU; Test type: Other; p = 0.789, Repeated measures analysis; Ratio = 1.031, 95% CI 2-sided [0.818 to 1.300]

9. Primary Outcome: Change From Baseline in Flow Cytometry: 6 Colour TBNK Panel- CD3+CD8+ and T Cell B Cell Natural Killer Lymphocytes (NKL)
Description: Whole blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Flow cytometry assessment included assessment of CD3+CD8+ and T Cell B Cell NKL. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Analysis was performed using repeated measures analysis adjusted for CD3+CD8+ and T Cell B Cell NKL log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: 10^9 cells/Liter
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
10^9 cells/Liter
  CD3+CD8+, Week 1, n=8, 25: number analyzed (Participants) | 8 | 25
  CD3+CD8+, Week 1, n=8, 25 | -0.041 (0.0390) | -0.005 (0.0222)
  CD3+CD8+, Week 4, n=8, 25: number analyzed (Participants) | 8 | 25
  CD3+CD8+, Week 4, n=8, 25 | 0.000 (0.0580) | -0.023 (0.0327)
  CD3+CD8+, Week 12, n=6, 25: number analyzed (Participants) | 6 | 25
  CD3+CD8+, Week 12, n=6, 25 | -0.056 (0.0418) | -0.037 (0.0215)
  CD3+CD8+, 12-Week FU, n=6, 21: number analyzed (Participants) | 6 | 21
  CD3+CD8+, 12-Week FU, n=6, 21 | -0.060 (0.0506) | -0.027 (0.0279)
  T Cell B Cell NKL, Week 1, n=8, 25: number analyzed (Participants) | 8 | 25
  T Cell B Cell NKL, Week 1, n=8, 25 | -0.123 (0.1557) | -0.020 (0.0881)
  T Cell B Cell NKL, Week 4, n=8, 25: number analyzed (Participants) | 8 | 25
  T Cell B Cell NKL, Week 4, n=8, 25 | 0.108 (0.2174) | -0.050 (0.1229)
  T Cell B Cell NKL, Week 12, n=6, 25: number analyzed (Participants) | 6 | 25
  T Cell B Cell NKL, Week 12, n=6, 25 | -0.093 (0.1792) | -0.006 (0.0925)
  T Cell B Cell NKL, 12-Week FU, n=6, 21: number analyzed (Participants) | 6 | 21
  T Cell B Cell NKL, 12-Week FU, n=6, 21 | -0.029 (0.2168) | -0.050 (0.1183)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD8+, Week 1; Test type: Other; p = 0.428, Repeated measures analysis; Mean Difference (Net) = 0.036, 95% CI 2-sided [-0.056 to 0.128]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD8+, Week 4; Test type: Other; p = 0.733, Repeated measures analysis; Mean Difference (Net) = -0.023, 95% CI 2-sided [-0.159 to 0.113]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD8+, Week 12; Test type: Other; p = 0.677, Repeated measures analysis; Mean Difference (Net) = 0.020, 95% CI 2-sided [-0.076 to 0.115]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD8+, 12-Week FU; Test type: Other; p = 0.569, Repeated measures analysis; Mean Difference (Net) = 0.033, 95% CI 2-sided [-0.084 to 0.151]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; T Cell B Cell NKL, Week 1; Test type: Other; p = 0.569, Repeated measures analysis; Mean Difference (Net) = 0.103, 95% CI 2-sided [-0.263 to 0.469]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; T Cell B Cell NKL, Week 4; Test type: Other; p = 0.534, Repeated measures analysis; Mean Difference (Net) = -0.157, 95% CI 2-sided [-0.668 to 0.354]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; T Cell B Cell NKL, Week 12; Test type: Other; p = 0.668, Repeated measures analysis; Mean Difference (Net) = 0.087, 95% CI 2-sided [-0.323 to 0.498]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; T Cell B Cell NKL, 12-Week FU; Test type: Other; p = 0.934, Repeated measures analysis; Mean Difference (Net) = -0.021, 95% CI 2-sided [-0.526 to 0.484]

10. Primary Outcome: Change From Baseline in Flow Cytometry: T Regulatory (Reg) Cell Foxp3- CD3+ CD4+, CD3+ CD8+ and CD3+
Description: Whole blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Flow cytometry assessment included assessment of CD3+ CD4+, CD3+ CD8+ and CD3+. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Analysis was performed using repeated measures analysis adjusted for CD3+ CD4+, CD3+ CD8+ and CD3+ Number of Cells (10^6/L) log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Ratio of T Reg cell
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of T Reg cell
  CD3+ CD4+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD3+ CD4+, Week 1, n=7, 23 | 0.905 (10.21) | 1.007 (5.65)
  CD3+ CD4+, Week 4, n=7, 22: number analyzed (Participants) | 7 | 22
  CD3+ CD4+, Week 4, n=7, 22 | 1.038 (11.31) | 0.976 (6.38)
  CD3+ CD4+, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD3+ CD4+, Week 12, n=5, 21 | 0.981 (10.55) | 1.004 (5.31)
  CD3+ CD4+, 12-Week FU, n=5, 17: number analyzed (Participants) | 5 | 17
  CD3+ CD4+, 12-Week FU, n=5, 17 | 0.926 (11.70) | 1.003 (6.39)
  CD3+ CD8+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD3+ CD8+, Week 1, n=7, 23 | 0.885 (9.97) | 0.983 (5.50)
  CD3+ CD8+, Week 4, n=7, 22: number analyzed (Participants) | 7 | 22
  CD3+ CD8+, Week 4, n=7, 22 | 0.981 (11.89) | 0.939 (6.66)
  CD3+ CD8+, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD3+ CD8+, Week 12, n=5, 21 | 0.878 (10.50) | 0.945 (5.40)
  CD3+ CD8+, 12-Week FU, n=5, 17: number analyzed (Participants) | 5 | 17
  CD3+ CD8+, 12-Week FU, n=5, 17 | 0.936 (10.99) | 0.965 (6.05)
  CD3+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD3+, Week 1, n=7, 23 | 0.901 (9.98) | 0.992 (5.54)
  CD3+, Week 4, n=7, 22: number analyzed (Participants) | 7 | 22
  CD3+, Week 4, n=7, 22 | 1.034 (12.99) | 0.938 (7.33)
  CD3+, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD3+, Week 12, n=5, 21 | 0.959 (9.62) | 0.993 (4.90)
  CD3+, 12-Week FU, n=5, 17: number analyzed (Participants) | 5 | 17
  CD3+, 12-Week FU, n=5, 17 | 0.944 (10.88) | 0.991 (6.00)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD4+, Week 1; Test type: Other; p = 0.369, Repeated measures analysis; Ratio = 1.112, 95% CI 2-sided [0.876 to 1.412]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD4+, Week 4; Test type: Other; p = 0.641, Repeated measures analysis; Ratio = 0.941, 95% CI 2-sided [0.721 to 1.228]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD4+, Week 12; Test type: Other; p = 0.844, Repeated measures analysis; Ratio = 1.024, 95% CI 2-sided [0.804 to 1.303]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD4+, 12-Week FU; Test type: Other; p = 0.558, Repeated measures analysis; Ratio = 1.082, 95% CI 2-sided [0.821 to 1.427]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD8+, Week 1; Test type: Other; p = 0.363, Repeated measures analysis; Ratio = 1.111, 95% CI 2-sided [0.880 to 1.402]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD8+, Week 4; Test type: Other; p = 0.751, Repeated measures analysis; Ratio = 0.957, 95% CI 2-sided [0.724 to 1.265]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD8+, Week 12; Test type: Other; p = 0.537, Repeated measures analysis; Ratio = 1.076, 95% CI 2-sided [0.846 to 1.370]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; CD3+ CD8+, 12-Week FU; Test type: Other; p = 0.806, Repeated measures analysis; Ratio = 1.032, 95% CI 2-sided [0.797 to 1.335]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; CD3+, Week 1; Test type: Other; p = 0.405, Repeated measures analysis; Ratio = 1.101, 95% CI 2-sided [0.872 to 1.391]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; CD3+, Week 4; Test type: Other; p = 0.519, Repeated measures analysis; Ratio = 0.907, 95% CI 2-sided [0.668 to 1.232]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; CD3+, Week 12; Test type: Other; p = 0.748, Repeated measures analysis; Ratio = 1.036, 95% CI 2-sided [0.831 to 1.291]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; CD3+, 12-Week FU; Test type: Other; p = 0.704, Repeated measures analysis; Ratio = 1.049, 95% CI 2-sided [0.811 to 1.356]

11. Primary Outcome: Change From Baseline in Flow Cytometry: T Reg Cell Foxp3: CD3+CD4+CD25+CD127-, CD3+CD4+foxP3+CD25+CD127-
Description: Whole blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Flow cytometry assessment included assessment of CD3+CD4+CD25+CD127- and CD3+CD4+foxP3+CD25+CD127-. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Analysis was performed using repeated measures analysis adjusted for CD3+CD4+CD25+CD127- and CD3+CD4+foxP3+CD25+CD127-Number of Cells (10^6 cells/L) log(Baseline value), treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/Liter
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
10^6 cells/Liter
  CD3+CD4+CD25+CD127-, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD3+CD4+CD25+CD127-, Week 1, n=7, 23 | -3.6 (8.35) | 2.9 (4.67)
  CD3+CD4+CD25+CD127-, Week 4, n=7, 22: number analyzed (Participants) | 7 | 22
  CD3+CD4+CD25+CD127-, Week 4, n=7, 22 | 1.4 (8.34) | -0.4 (4.70)
  CD3+CD4+CD25+CD127-, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD3+CD4+CD25+CD127-, Week 12, n=5, 21 | -9.4 (9.87) | -3.1 (4.94)
  CD3+CD4+CD25+CD127-, 12-Week FU, n=5, 17: number analyzed (Participants) | 5 | 17
  CD3+CD4+CD25+CD127-, 12-Week FU, n=5, 17 | -12.9 (9.92) | -2.3 (5.43)
  CD3+CD4+foxP3+CD25+CD127, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD3+CD4+foxP3+CD25+CD127, Week 1, n=7, 23 | 0.8 (6.39) | 2.8 (3.58)
  CD3+CD4+foxP3+CD25+CD127, Week 4, n=7, 22: number analyzed (Participants) | 7 | 22
  CD3+CD4+foxP3+CD25+CD127, Week 4, n=7, 22 | 4.3 (7.05) | 2.0 (3.98)
  CD3+CD4+foxP3+CD25+CD127, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD3+CD4+foxP3+CD25+CD127, Week 12, n=5, 21 | 2.7 (7.99) | -4.4 (3.91)
  CD3+CD4+foxP3+CD25+CD127,12-Week FU, n=5,17: number analyzed (Participants) | 5 | 17
  CD3+CD4+foxP3+CD25+CD127,12-Week FU, n=5,17 | -8.7 (5.94) | -4.6 (3.15)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+CD25+CD127-, Week 1; Test type: Other; p = 0.501, Repeated measures analysis; Mean Difference (Net) = 6.5, 95% CI 2-sided [-13.1 to 26.1]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+CD25+CD127-, Week 4; Test type: Other; p = 0.852, Repeated measures analysis; Mean Difference (Net) = -1.8, 95% CI 2-sided [-21.6 to 18.0]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+CD25+CD127-, Week 12; Test type: Other; p = 0.572, Repeated measures analysis; Mean Difference (Net) = 6.3, 95% CI 2-sided [-16.4 to 29.0]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+CD25+CD127-, 12-Week FU; Test type: Other; p = 0.363, Repeated measures analysis; Mean Difference (Net) = 10.5, 95% CI 2-sided [-13.0 to 34.1]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+foxP3+CD25+CD127-, Week 1; Test type: Other; p = 0.788, Repeated measures analysis; Mean Difference (Net) = 2.0, 95% CI 2-sided [-13.0 to 17.0]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+foxP3+CD25+CD127-, Week 4; Test type: Other; p = 0.786, Repeated measures analysis; Mean Difference (Net) = -2.2, 95% CI 2-sided [-18.8 to 14.4]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+foxP3+CD25+CD127-, Week 12; Test type: Other; p = 0.433, Repeated measures analysis; Mean Difference (Net) = -7.1, 95% CI 2-sided [-25.4 to 11.2]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; CD3+CD4+foxP3+CD25+CD127-, 12-Week FU; Test type: Other; p = 0.550, Repeated measures analysis; Mean Difference (Net) = 4.1, 95% CI 2-sided [-9.8 to 18.0]

12. Primary Outcome: Change From Baseline in T Helper Cell Panel Events
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. T Helper Cell Panel included analysis of CD45+3+8-4+CCR6+CXCR3+38+DR+, CD45+3+8-4+CCR6+CXCR3-38+DR+, CD45+3+8-4+CCR6-CXCR3+38+DR+, CD45+3+8-4+CCR6-CXCR3-38+DR+, CD45+CD3+CD8-CD4+, CD45+CD3+CD8-CD4+CCR6+CXCR3+, CD45+CD3+CD8-CD4+CCR6+CXCR3-, CD45+CD3+CD8-CD4+CCR6-CXCR3+ and CD45+CD3+CD8-CD4+CCR6-CXCR3-. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Analysis was performed using repeated measures analysis adjusted for T Helper Cell Panel Events (EVENTS) Baseline value, treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Events
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Events
  CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 1, n=7, 23 | -48.6 (13.50) | -34.0 (7.35)
  CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 4, n=7, 21 | -14.5 (18.36) | -6.1 (10.63)
  CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 12, n=5, 22 | 42.3 (37.80) | -6.9 (17.69)
  CD45+3+8-4+CCR6+CXCR3+38+DR+,12-Week FU,n=5,18: number analyzed (Participants) | 5 | 18
  CD45+3+8-4+CCR6+CXCR3+38+DR+,12-Week FU,n=5,18 | 11.5 (16.47) | -18.7 (8.66)
  CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 1, n=7, 23 | -17.0 (6.80) | -10.5 (3.62)
  CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 4, n=7, 21 | 14.2 (15.65) | 12.2 (9.10)
  CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 12, n=5, 22 | 3.4 (16.09) | -3.0 (7.55)
  CD45+3+8-4+CCR6+CXCR3-38+DR+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+3+8-4+CCR6+CXCR3-38+DR+, 12-Week FU, n=5, 18 | 8.9 (12.29) | 3.3 (6.36)
  CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 1, n=7, 23 | -73.2 (82.46) | -129.2 (46.04)
  CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 4, n=7, 21 | -159.6 (60.51) | -108.0 (35.05)
  CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 12, n=5, 22 | 219.2 (299.65) | 77.7 (146.73)
  CD45+3+8-4+CCR6-CXCR3+38+DR+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+3+8-4+CCR6-CXCR3+38+DR+, 12-Week FU, n=5, 18 | 33.9 (66.09) | -104.0 (34.73)
  CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 1, n=7, 23 | -70.9 (25.90) | -70.5 (14.03)
  CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 4, n=7, 21 | -38.9 (30.69) | -56.3 (17.93)
  CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 12, n=5, 22 | -16.4 (198.13) | 43.0 (92.38)
  CD45+3+8-4+CCR6-CXCR3-38+DR+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+3+8-4+CCR6-CXCR3-38+DR+, 12-Week FU, n=5, 18 | -12.7 (33.50) | -59.9 (17.32)
  CD45+CD3+CD8-CD4+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+CD3+CD8-CD4+, Week 1, n=7, 23 | -3845.3 (2648.60) | -163.0 (1444.61)
  CD45+CD3+CD8-CD4+, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+CD3+CD8-CD4+, Week 4, n=7, 21 | 1622.8 (2973.60) | 1075.1 (1723.09)
  vCD45+CD3+CD8-CD4+, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  vCD45+CD3+CD8-CD4+, Week 12, n=5, 22 | 2112.9 (4211.63) | 1006.9 (2026.47)
  CD45+CD3+CD8-CD4+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+CD3+CD8-CD4+, 12-Week FU, n=5, 18 | 1799.0 (2589.05) | -1832.0 (1366.65)
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 1, n=7, 23 | -514.6 (647.85) | -1030.2 (345.07)
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 4, n=7, 21 | -116.6 (757.58) | -316.5 (438.76)
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 12, n=5, 22 | -252.9 (827.53) | -506.4 (389.97)
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+CD3+CD8-CD4+CCR6+CXCR3+, 12-Week FU, n=5, 18 | -688.1 (792.26) | -463.0 (412.22)
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 1, n=7, 23 | -817.1 (393.10) | -654.5 (212.18)
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 4, n=7, 21 | 197.7 (475.88) | 14.2 (277.06)
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 12, n=5, 22 | 48.8 (541.14) | -219.7 (253.92)
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+CD3+CD8-CD4+CCR6+CXCR3-, 12-Week FU, n=5, 18 | -311.6 (553.32) | -509.2 (291.09)
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 1, n=7, 23 | 371.8 (1026.17) | 1521.8 (547.18)
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 4, n=7, 21 | -24.5 (1678.23) | -292.5 (967.00)
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 12, n=5, 22 | 2790.5 (2510.67) | 1443.1 (1209.66)
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+CD3+CD8-CD4+CCR6-CXCR3+, 12-Week FU, n=5, 18 | 2295.9 (1787.02) | 607.0 (927.11)
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 1, n=7, 23: number analyzed (Participants) | 7 | 23
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 1, n=7, 23 | -3231.4 (2162.58) | 45.4 (1187.37)
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 4, n=7, 21: number analyzed (Participants) | 7 | 21
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 4, n=7, 21 | 2084.9 (2873.95) | 1637.6 (1665.46)
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 12, n=5, 22: number analyzed (Participants) | 5 | 22
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 12, n=5, 22 | -1273.9 (2413.90) | 161.4 (1209.82)
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD45+CD3+CD8-CD4+CCR6-CXCR3-, 12-Week FU, n=5, 18 | -106.6 (1690.64) | -1316.7 (892.55)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 1; Test type: Other; p = 0.350, Repeated measures analysis; Mean Difference (Net) = 14.6, 95% CI 2-sided [-16.9 to 46.1]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 4; Test type: Other; p = 0.697, Repeated measures analysis; Mean Difference (Net) = 8.4, 95% CI 2-sided [-35.3 to 52.0]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3+38+DR+, Week 12; Test type: Other; p = 0.249, Repeated measures analysis; Mean Difference (Net) = -49.2, 95% CI 2-sided [-135.2 to 36.8]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3+38+DR+, 12-Week FU; Test type: Other; p = 0.119, Repeated measures analysis; Mean Difference (Net) = -30.1, 95% CI 2-sided [-68.6 to 8.3]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 1; Test type: Other; p = 0.403, Repeated measures analysis; Mean Difference (Net) = 6.5, 95% CI 2-sided [-9.3 to 22.4]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 4; Test type: Other; p = 0.910, Repeated measures analysis; Mean Difference (Net) = -2.1, 95% CI 2-sided [-39.4 to 35.2]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3-38+DR+, Week 12; Test type: Other; p = 0.718, Repeated measures analysis; Mean Difference (Net) = -6.5, 95% CI 2-sided [-43.1 to 30.1]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6+CXCR3-38+DR+, 12-Week FU; Test type: Other; p = 0.687, Repeated measures analysis; Mean Difference (Net) = -5.7, 95% CI 2-sided [-34.4 to 23.0]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 1; Test type: Other; p = 0.559, Repeated measures analysis; Mean Difference (Net) = -56.0, 95% CI 2-sided [-249.8 to 137.7]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 4; Test type: Other; p = 0.470, Repeated measures analysis; Mean Difference (Net) = 51.6, 95% CI 2-sided [-93.9 to 197.0]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3+38+DR+, Week 12; Test type: Other; p = 0.675, Repeated measures analysis; Mean Difference (Net) = -141.5, 95% CI 2-sided [-829.2 to 546.3]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3+38+DR+, 12-Week FU; Test type: Other; p = 0.080, Repeated measures analysis; Mean Difference (Net) = -137.9, 95% CI 2-sided [-294.0 to 18.2]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 1; Test type: Other; p = 0.989, Repeated measures analysis; Mean Difference (Net) = 0.4, 95% CI 2-sided [-60.5 to 61.3]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 4; Test type: Other; p = 0.634, Repeated measures analysis; Mean Difference (Net) = -17.4, 95% CI 2-sided [-94.3 to 59.6]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3-38+DR+, Week 12; Test type: Other; p = 0.789, Repeated measures analysis; Mean Difference (Net) = 59.4, 95% CI 2-sided [-395.2 to 513.9]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 180 mg; CD45+3+8-4+CCR6-CXCR3-38+DR+, 12-Week FU; Test type: Other; p = 0.249, Repeated measures analysis; Mean Difference (Net) = -47.2, 95% CI 2-sided [-135.5 to 41.0]
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+, Week 1; Test type: Other; p = 0.234, Repeated measures analysis; Mean Difference (Net) = 3682.3, 95% CI 2-sided [-2511.9 to 9876.5]
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+, Week 4; Test type: Other; p = 0.875, Repeated measures analysis; Mean Difference (Net) = -547.6, 95% CI 2-sided [-7612.6 to 6517.3]
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+, Week 12; Test type: Other; p = 0.815, Repeated measures analysis; Mean Difference (Net) = -1106.0, 95% CI 2-sided [-10706.0 to 8494.1]
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+, 12-Week FU; Test type: Other; p = 0.230, Repeated measures analysis; Mean Difference (Net) = -3631.0, 95% CI 2-sided [-9738.9 to 2476.8]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 1; Test type: Other; p = 0.489, Repeated measures analysis; Mean Difference (Net) = -515.6, 95% CI 2-sided [-2021.4 to 990.1]
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 4; Test type: Other; p = 0.822, Repeated measures analysis; Mean Difference (Net) = -199.8, 95% CI 2-sided [-2001.7 to 1602.0]
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3+, Week 12; Test type: Other; p = 0.784, Repeated measures analysis; Mean Difference (Net) = -253.5, 95% CI 2-sided [-2136.7 to 1629.7]
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3+, 12-Week FU; Test type: Other; p = 0.804, Repeated measures analysis; Mean Difference (Net) = 225.1, 95% CI 2-sided [-1633.1 to 2083.2]
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 1; Test type: Other; p = 0.719, Repeated measures analysis; Mean Difference (Net) = 162.7, 95% CI 2-sided [-754.5 to 1079.9]
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 4; Test type: Other; p = 0.742, Repeated measures analysis; Mean Difference (Net) = -183.5, 95% CI 2-sided [-1317.4 to 950.3]
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3-, Week 12; Test type: Other; p = 0.658, Repeated measures analysis; Mean Difference (Net) = -268.5, 95% CI 2-sided [-1507.5 to 970.5]
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6+CXCR3-, 12-Week FU; Test type: Other; p = 0.755, Repeated measures analysis; Mean Difference (Net) = -197.6, 95% CI 2-sided [-1499.3 to 1104.2]
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 1; Test type: Other; p = 0.333, Repeated measures analysis; Mean Difference (Net) = 1150.0, 95% CI 2-sided [-1250.0 to 3550.0]
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 4; Test type: Other; p = 0.891, Repeated measures analysis; Mean Difference (Net) = -268.0, 95% CI 2-sided [-4269.2 to 3733.3]
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3+, Week 12; Test type: Other; p = 0.633, Repeated measures analysis; Mean Difference (Net) = -1347.4, 95% CI 2-sided [-7073.1 to 4378.3]
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3+, 12-Week FU; Test type: Other; p = 0.410, Repeated measures analysis; Mean Difference (Net) = -1688.9, 95% CI 2-sided [-5864.1 to 2486.2]
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 1; Test type: Other; p = 0.196, Repeated measures analysis; Mean Difference (Net) = 3276.8, 95% CI 2-sided [-1786.0 to 8339.6]
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 4; Test type: Other; p = 0.894, Repeated measures analysis; Mean Difference (Net) = -447.3, 95% CI 2-sided [-7285.5 to 6390.8]
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3-, Week 12; Test type: Other; p = 0.600, Repeated measures analysis; Mean Difference (Net) = 1435.3, 95% CI 2-sided [-4101.4 to 6972.0]
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 180 mg; CD45+CD3+CD8-CD4+CCR6-CXCR3-, 12-Week FU; Test type: Other; p = 0.534, Repeated measures analysis; Mean Difference (Net) = -1210.2, 95% CI 2-sided [-5213.1 to 2792.7]

13. Primary Outcome: Change From Baseline in Flow Cytometry: CD16+ Monocyte Panel: CD14-HLA-DR+CD11cbr+CD123-, CD14br+CD16+, CD14br+CD16-, CD14lo+CD16br+
Description: Whole blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Flow cytometry assessment included assessment of CD14-HLA-DR+CD11cbr+CD123-, CD14br+CD16+, CD14br+CD16- and CD14lo+CD16br+. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Analysis was performed using repeated measures analysis adjusted for CD14-HLA-DR+CD11cbr+CD123-, CD14br+CD16+, CD14br+CD16- and CD14lo+CD16br+ (10^3/Liter) baseline value, treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: 10^3 cells/Liter
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
10^3 cells/Liter
  CD14-HLA-DR+CD11cbr+CD123-, Week 1, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14-HLA-DR+CD11cbr+CD123-, Week 1, n=5, 18 | -2017.6 (2452.91) | 738.7 (1266.25)
  CD14-HLA-DR+CD11cbr+CD123-, Week 4, n=6, 22: number analyzed (Participants) | 6 | 22
  CD14-HLA-DR+CD11cbr+CD123-, Week 4, n=6, 22 | 2766.3 (3220.54) | 2278.8 (1696.12)
  CD14-HLA-DR+CD11cbr+CD123-, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD14-HLA-DR+CD11cbr+CD123-, Week 12, n=5, 21 | 5730.4 (5085.86) | 5453.0 (2399.11)
  CD14-HLA-DR+CD11cbr+CD123-, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14-HLA-DR+CD11cbr+CD123-, 12-Week FU, n=5, 18 | 5785.6 (5081.59) | 5474.0 (2439.59)
  CD14br+CD16+, Week 1, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14br+CD16+, Week 1, n=5, 18 | -5376.0 (4748.95) | 1491.0 (2452.69)
  CD14br+CD16+, Week 4, n=6, 22: number analyzed (Participants) | 6 | 22
  CD14br+CD16+, Week 4, n=6, 22 | -5635.3 (5971.99) | 2724.3 (3117.17)
  CD14br+CD16+, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD14br+CD16+, Week 12, n=5, 21 | 25351.6 (9433.73) | 2668.0 (4589.28)
  CD14br+CD16+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14br+CD16+, 12-Week FU, n=5, 18 | 8557.2 (9914.93) | 4800.0 (5266.23)
  CD14br+CD16-, Week 1, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14br+CD16-, Week 1, n=5, 18 | 40079.7 (40456.86) | 17662.7 (21211.91)
  CD14br+CD16-, Week 4, n=6, 22: number analyzed (Participants) | 6 | 22
  CD14br+CD16-, Week 4, n=6, 22 | -17173.8 (24181.15) | 10485.9 (12635.98)
  CD14br+CD16-, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD14br+CD16-, Week 12, n=5, 21 | -2981.8 (37788.70) | 13201.2 (18684.22)
  CD14br+CD16-, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14br+CD16-, 12-Week FU, n=5, 18 | 31906.6 (45766.70) | -31512.8 (24027.16)
  CD14lo+CD16br+, Week 1, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14lo+CD16br+, Week 1, n=5, 18 | 11248.2 (6598.36) | 4334.6 (3466.71)
  CD14lo+CD16br+, Week 4, n=6, 22: number analyzed (Participants) | 6 | 22
  CD14lo+CD16br+, Week 4, n=6, 22 | 2522.9 (3757.96) | 291.3 (1959.54)
  CD14lo+CD16br+, Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  CD14lo+CD16br+, Week 12, n=5, 21 | 10938.4 (5088.36) | 759.2 (2534.27)
  CD14lo+CD16br+, 12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  CD14lo+CD16br+, 12-Week FU, n=5, 18 | 24737.0 (7758.65) | 3992.8 (4134.52)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; CD14-HLA-DR+CD11cbr+CD123-, Week 1; Test type: Other; p = 0.328, Repeated measures analysis; Mean Difference (Net) = 2756.3, 95% CI 2-sided [-2953.7 to 8466.3]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; CD14-HLA-DR+CD11cbr+CD123-, Week 4; Test type: Other; p = 0.895, Repeated measures analysis; Mean Difference (Net) = -487.5, 95% CI 2-sided [-8003.7 to 7028.6]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; CD14-HLA-DR+CD11cbr+CD123-, Week 12; Test type: Other; p = 0.961, Repeated measures analysis; Mean Difference (Net) = -277.4, 95% CI 2-sided [-12001.0 to 11446.2]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; CD14-HLA-DR+CD11cbr+CD123-, 12-Week FU; Test type: Other; p = 0.956, Repeated measures analysis; Mean Difference (Net) = -311.6, 95% CI 2-sided [-11960.5 to 11337.4]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16+, Week 1; Test type: Other; p = 0.212, Repeated measures analysis; Mean Difference (Net) = 6866.9, 95% CI 2-sided [-4230.7 to 17964.6]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16+, Week 4; Test type: Other; p = 0.227, Repeated measures analysis; Mean Difference (Net) = 8359.6, 95% CI 2-sided [-5533.3 to 22252.5]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16+, Week 12; Test type: Other; p = 0.040, Repeated measures analysis; Mean Difference (Net) = -22683.6, 95% CI 2-sided [-44298.5 to -1068.8]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16+, 12-Week FU; Test type: Other; p = 0.741, Repeated measures analysis; Mean Difference (Net) = -3757.2, 95% CI 2-sided [-27146.0 to 19631.6]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16-, Week 1; Test type: Other; p = 0.628, Repeated measures analysis; Mean Difference (Net) = -22417.0, 95% CI 2-sided [-116677.8 to 71843.8]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16-, Week 4; Test type: Other; p = 0.321, Repeated measures analysis; Mean Difference (Net) = 27659.7, 95% CI 2-sided [-28567.8 to 83887.1]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16-, Week 12; Test type: Other; p = 0.704, Repeated measures analysis; Mean Difference (Net) = 16182.9, 95% CI 2-sided [-70377.0 to 102742.9]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; CD14br+CD16-, 12-Week FU; Test type: Other; p = 0.232, Repeated measures analysis; Mean Difference (Net) = -63419.4, 95% CI 2-sided [-170364.9 to 43526.1]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; CD14lo+CD16br+, Week 1; Test type: Other; p = 0.366, Repeated measures analysis; Mean Difference (Net) = -6913.6, 95% CI 2-sided [-22588.4 to 8761.1]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; CD14lo+CD16br+, Week 4; Test type: Other; p = 0.603, Repeated measures analysis; Mean Difference (Net) = -2231.6, 95% CI 2-sided [-10976.8 to 6513.6]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; CD14lo+CD16br+, Week 12; Test type: Other; p = 0.084, Repeated measures analysis; Mean Difference (Net) = -10179.1, 95% CI 2-sided [-21827.4 to 1469.2]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 180 mg; CD14lo+CD16br+, 12-Week FU; Test type: Other; p = 0.026, Repeated measures analysis; Mean Difference (Net) = -20744.2, 95% CI 2-sided [-38771.8 to -2716.5]

14. Primary Outcome: Change From Baseline in Flow Cytometry: CD16+ Monocyte Panel: CD14-CD16+CD66b+
Description: Whole blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Flow cytometry assessment included assessment of CD14-CD16+CD66b+ cell. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Analysis was performed using repeated measures analysis adjusted for CD14-CD16+CD66b+ (10^6/Liter) baseline value, treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/Liter
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
10^6 cells/Liter
  Week 1, n=5, 19: number analyzed (Participants) | 5 | 19
  Week 1, n=5, 19 | -559.0 (269.84) | -380.9 (137.31)
  Week 4, n=6, 22: number analyzed (Participants) | 6 | 22
  Week 4, n=6, 22 | -581.9 (377.03) | -41.5 (196.72)
  Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  Week 12, n=5, 21 | -125.9 (460.53) | -378.6 (229.47)
  12-Week FU, n=5, 18: number analyzed (Participants) | 5 | 18
  12-Week FU, n=5, 18 | -240.9 (430.65) | -199.3 (219.73)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Week 1; Test type: Other; p = 0.564, Repeated measures analysis; Mean Difference (Net) = 178.2, 95% CI 2-sided [-448.3 to 804.6]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Week 4; Test type: Other; p = 0.216, Repeated measures analysis; Mean Difference (Net) = 540.4, 95% CI 2-sided [-335.7 to 1416.5]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; Week 12; Test type: Other; p = 0.629, Repeated measures analysis; Mean Difference (Net) = -252.6, 95% CI 2-sided [-1326.0 to 820.8]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU; Test type: Other; p = 0.932, Repeated measures analysis; Mean Difference (Net) = 41.6, 95% CI 2-sided [-962.2 to 1045.5]

15. Primary Outcome: Change From Baseline in Complement Biomarkers: Complement Component 3 (C3), Complement Component 4 (C4)
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Complement biomarkers included analysis of Complement C3 and Complement C4. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of complement biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of complement biomarker
  Complement C3, Week 1, n=9, 25: number analyzed (Participants) | 9 | 25
  Complement C3, Week 1, n=9, 25 | 0.967 (7.43) | 0.982 (11.76)
  Complement C3, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Complement C3, Week 2, n=8, 26 | 0.957 (11.72) | 0.963 (14.15)
  Complement C3, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement C3, Week 4, n=9, 27 | 1.045 (18.42) | 0.959 (12.62)
  Complement C3, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Complement C3, Week 6, n=7, 27 | 1.060 (12.00) | 0.991 (11.71)
  Complement C3, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Complement C3, Week 8, n=7, 25 | 1.021 (12.54) | 1.009 (10.85)
  Complement C3, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Complement C3, Week 12, n=7, 24 | 0.988 (9.37) | 1.003 (11.34)
  Complement C3, 12-Week FU, n=7, 22: number analyzed (Participants) | 7 | 22
  Complement C3, 12-Week FU, n=7, 22 | 1.005 (19.15) | 0.995 (10.65)
  Complement C4, Week 1, n=9, 25: number analyzed (Participants) | 9 | 25
  Complement C4, Week 1, n=9, 25 | 1.005 (11.40) | 0.969 (13.13)
  Complement C4, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Complement C4, Week 2, n=8, 26 | 0.949 (9.64) | 0.984 (16.45)
  Complement C4, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement C4, Week 4, n=9, 27 | 0.999 (12.06) | 0.945 (14.63)
  Complement C4, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Complement C4, Week 6, n=7, 27 | 0.990 (10.31) | 0.985 (17.32)
  Complement C4, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Complement C4, Week 8, n=7, 25 | 0.979 (7.66) | 1.006 (13.53)
  Complement C4, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Complement C4, Week 12, n=7, 24 | 0.942 (15.57) | 0.994 (12.75)
  Complement C4, 12-Week FU, n=7, 22: number analyzed (Participants) | 7 | 22
  Complement C4, 12-Week FU, n=7, 22 | 0.982 (12.88) | 0.986 (14.72)

16. Primary Outcome: Change From Baseline in Complement Biomarkers: Complement Component 4a (C4a), Complement Component 5a (C5a), Complement Split Factor SC5b-9, Soluble Cluster of Differentiation 163 (sCD163)
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Complement biomarkers included analysis of Complement C4a, Complement C5a, Complement Split Factor SC5b-9 and Soluble CD163. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of complement biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of complement biomarker
  Complement C4a, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement C4a, Week 1, n=9, 27 | 1.159 (115.81) | 0.990 (67.63)
  Complement C4a, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Complement C4a, Week 2, n=8, 26 | 0.881 (55.58) | 1.156 (75.77)
  Complement C4a, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement C4a, Week 4, n=9, 27 | 0.840 (40.85) | 1.100 (46.87)
  Complement C4a, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Complement C4a, Week 6, n=7, 27 | 0.914 (66.71) | 0.860 (53.87)
  Complement C4a, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Complement C4a, Week 8, n=7, 25 | 1.017 (44.16) | 0.998 (60.41)
  Complement C4a, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Complement C4a, Week 12, n=7, 24 | 0.927 (58.05) | 0.901 (93.48)
  Complement C4a, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Complement C4a, 12-Week FU, n=7, 21 | 1.104 (40.27) | 1.221 (56.53)
  Complement C5a, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement C5a, Week 1, n=9, 27 | 0.927 (19.42) | 0.991 (29.67)
  Complement C5a, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Complement C5a, Week 2, n=8, 26 | 1.154 (36.82) | 1.015 (55.60)
  Complement C5a, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement C5a, Week 4, n=9, 27 | 0.943 (16.76) | 1.010 (35.63)
  Complement C5a, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Complement C5a, Week 6, n=7, 27 | 1.139 (61.77) | 1.044 (33.94)
  Complement C5a, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Complement C5a, Week 8, n=7, 25 | 0.980 (13.71) | 0.957 (26.95)
  Complement C5a, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Complement C5a, Week 12, n=7, 24 | 1.012 (8.41) | 0.995 (29.49)
  Complement C5a, 12-Week FU, n=7, 22: number analyzed (Participants) | 7 | 22
  Complement C5a, 12-Week FU, n=7, 22 | 1.152 (42.75) | 1.130 (32.16)
  Complement Split Factor SC5b-9, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement Split Factor SC5b-9, Week 1, n=9, 27 | 0.971 (37.46) | 1.020 (43.70)
  Complement Split Factor SC5b-9, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Complement Split Factor SC5b-9, Week 2, n=8, 26 | 1.078 (28.80) | 1.040 (60.64)
  Complement Split Factor SC5b-9, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Complement Split Factor SC5b-9, Week 4, n=9, 27 | 0.930 (43.01) | 1.126 (41.04)
  Complement Split Factor SC5b-9, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Complement Split Factor SC5b-9, Week 6, n=7, 27 | 0.989 (23.18) | 1.084 (53.90)
  Complement Split Factor SC5b-9, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Complement Split Factor SC5b-9, Week 8, n=7, 25 | 0.889 (35.48) | 1.055 (67.53)
  Complement Split Factor SC5b-9, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Complement Split Factor SC5b-9, Week 12, n=7, 24 | 0.883 (30.26) | 0.843 (72.14)
  Complement Split Factor SC5b-9,12-Week FU, n=7, 22: number analyzed (Participants) | 7 | 22
  Complement Split Factor SC5b-9,12-Week FU, n=7, 22 | 1.039 (69.05) | 1.041 (38.60)
  sCD163, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  sCD163, Week 1, n=9, 27 | 0.993 (24.28) | 0.963 (16.38)
  sCD163, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  sCD163, Week 2, n=8, 26 | 1.101 (17.80) | 0.954 (17.14)
  sCD163, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  sCD163, Week 4, n=9, 27 | 0.986 (15.89) | 0.947 (27.10)
  sCD163, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  sCD163, Week 6, n=7, 27 | 0.938 (20.83) | 0.959 (30.14)
  sCD163, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  sCD163, Week 8, n=7, 25 | 0.938 (30.03) | 0.950 (28.73)
  sCD163, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  sCD163, Week 12, n=7, 24 | 0.937 (24.86) | 0.915 (35.29)
  sCD163, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  sCD163, 12-Week FU, n=7, 21 | 1.200 (32.94) | 0.994 (28.84)

17. Primary Outcome: Change From Baseline in Mechanistic Biomarkers
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Mechanistic biomarkers included analysis of Interleukin 1 Beta, Interleukin 10, Interleukin 15, Interleukin 17 Alpha, Interleukin 17F, Interleukin 8 and Tumor Necrosis Factor. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. NA indicates that data is not available since 100% of the data was below limit of quantification at all time points. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of mechanistic biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of mechanistic biomarker
  Interleukin 1 Beta, Week 1, n=9, 26: number analyzed (Participants) | 9 | 26
  Interleukin 1 Beta, Week 1, n=9, 26 | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability. | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability.
  Interleukin 1 Beta, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Interleukin 1 Beta, Week 2, n=8, 26 | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability. | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability.
  Interleukin 1 Beta, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Interleukin 1 Beta, Week 4, n=9, 27 | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability. | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability.
  Interleukin 1 Beta, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Interleukin 1 Beta, Week 6, n=7, 27 | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability. | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability.
  Interleukin 1 Beta, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Interleukin 1 Beta, Week 8, n=7, 25 | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability. | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability.
  Interleukin 1 Beta, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Interleukin 1 Beta, Week 12, n=7, 24 | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability. | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability.
  Interleukin 1 Beta, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Interleukin 1 Beta, 12-Week FU, n=7, 21 | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability. | 1.000 (NA) — 100% of data was below limit of quantification at all time points, hence no variability.
  Interleukin 10, Week 1, n=9, 26: number analyzed (Participants) | 9 | 26
  Interleukin 10, Week 1, n=9, 26 | 0.962 (11.55) | 0.994 (28.47)
  Interleukin 10, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Interleukin 10, Week 2, n=8, 26 | 1.206 (45.35) | 1.048 (37.27)
  Interleukin 10, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Interleukin 10, Week 4, n=9, 27 | 0.875 (41.69) | 0.985 (32.52)
  Interleukin 10, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Interleukin 10, Week 6, n=7, 27 | 0.842 (47.84) | 0.960 (17.66)
  Interleukin 10, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Interleukin 10, Week 8, n=7, 25 | 1.197 (50.41) | 0.969 (30.23)
  Interleukin 10, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Interleukin 10, Week 12, n=7, 24 | 0.842 (47.84) | 0.989 (21.36)
  Interleukin 10, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Interleukin 10, 12-Week FU, n=7, 21 | 0.842 (47.84) | 1.230 (62.91)
  Interleukin 15, Week 1, n=9, 27: number analyzed (Participants) | 9 | 27
  Interleukin 15, Week 1, n=9, 27 | 1.001 (12.70) | 0.950 (59.23)
  Interleukin 15, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Interleukin 15, Week 2, n=8, 26 | 0.882 (41.99) | 0.849 (102.76)
  Interleukin 15, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Interleukin 15, Week 4, n=9, 27 | 1.206 (47.87) | 0.831 (84.07)
  Interleukin 15, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Interleukin 15, Week 6, n=7, 27 | 1.297 (48.81) | 0.904 (90.53)
  Interleukin 15, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Interleukin 15, Week 8, n=7, 25 | 0.871 (37.95) | 0.865 (90.30)
  Interleukin 15, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Interleukin 15, Week 12, n=7, 24 | 0.871 (37.95) | 0.771 (82.21)
  Interleukin 15, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Interleukin 15, 12-Week FU, n=7, 21 | 0.871 (37.95) | 0.636 (111.86)
  Interleukin 17 Alpha, Week 1, n=9, 25: number analyzed (Participants) | 9 | 25
  Interleukin 17 Alpha, Week 1, n=9, 25 | 0.806 (53.03) | 1.054 (93.04)
  Interleukin 17 Alpha, Week 2, n=8, 25: number analyzed (Participants) | 8 | 25
  Interleukin 17 Alpha, Week 2, n=8, 25 | 0.935 (75.58) | 0.942 (72.24)
  Interleukin 17 Alpha, Week 4, n=9, 26: number analyzed (Participants) | 9 | 26
  Interleukin 17 Alpha, Week 4, n=9, 26 | 0.995 (91.45) | 0.911 (102.66)
  Interleukin 17 Alpha, Week 6, n=7, 26: number analyzed (Participants) | 7 | 26
  Interleukin 17 Alpha, Week 6, n=7, 26 | 1.015 (76.60) | 0.867 (90.15)
  Interleukin 17 Alpha, Week 8, n=7, 23: number analyzed (Participants) | 7 | 23
  Interleukin 17 Alpha, Week 8, n=7, 23 | 0.905 (77.24) | 1.005 (135.76)
  Interleukin 17 Alpha, Week 12, n=7, 23: number analyzed (Participants) | 7 | 23
  Interleukin 17 Alpha, Week 12, n=7, 23 | 1.007 (87.84) | 0.857 (101.45)
  Interleukin 17 Alpha, 12-Week FU, n=7, 20: number analyzed (Participants) | 7 | 20
  Interleukin 17 Alpha, 12-Week FU, n=7, 20 | 0.969 (155.67) | 0.999 (150.12)
  Interleukin 17F, Week 1, n=9, 25: number analyzed (Participants) | 9 | 25
  Interleukin 17F, Week 1, n=9, 25 | 1.153 (36.21) | 0.797 (78.96)
  Interleukin 17F, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Interleukin 17F, Week 2, n=8, 26 | 1.062 (74.38) | 0.911 (72.36)
  Interleukin 17F, Week 4, n=9, 26: number analyzed (Participants) | 9 | 26
  Interleukin 17F, Week 4, n=9, 26 | 0.966 (21.09) | 0.948 (89.47)
  Interleukin 17F, Week 6, n=7, 25: number analyzed (Participants) | 7 | 25
  Interleukin 17F, Week 6, n=7, 25 | 0.787 (32.55) | 1.013 (107.49)
  Interleukin 17F, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Interleukin 17F, Week 8, n=7, 25 | 0.947 (19.20) | 0.815 (91.93)
  Interleukin 17F, Week 12, n=7, 23: number analyzed (Participants) | 7 | 23
  Interleukin 17F, Week 12, n=7, 23 | 1.002 (74.09) | 0.884 (100.03)
  Interleukin 17F, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Interleukin 17F, 12-Week FU, n=7, 21 | 1.130 (101.51) | 0.741 (90.62)
  Interleukin 8, Week 1, n=9, 26: number analyzed (Participants) | 9 | 26
  Interleukin 8, Week 1, n=9, 26 | 1.104 (40.98) | 1.081 (74.78)
  Interleukin 8, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Interleukin 8, Week 2, n=8, 26 | 1.505 (43.78) | 0.861 (78.64)
  Interleukin 8, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Interleukin 8, Week 4, n=9, 27 | 1.102 (38.30) | 0.773 (82.48)
  Interleukin 8, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Interleukin 8, Week 6, n=7, 27 | 1.229 (61.82) | 0.720 (72.70)
  Interleukin 8, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Interleukin 8, Week 8, n=7, 25 | 1.547 (53.88) | 0.761 (80.51)
  Interleukin 8, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Interleukin 8, Week 12, n=7, 24 | 1.240 (49.03) | 0.850 (80.98)
  Interleukin 8, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Interleukin 8, 12-Week FU, n=7, 21 | 1.191 (42.58) | 0.841 (96.92)
  Tumor Necrosis Factor, Week 1, n=9, 26: number analyzed (Participants) | 9 | 26
  Tumor Necrosis Factor, Week 1, n=9, 26 | 0.976 (15.20) | 0.994 (18.45)
  Tumor Necrosis Factor, Week 2, n=8, 26: number analyzed (Participants) | 8 | 26
  Tumor Necrosis Factor, Week 2, n=8, 26 | 0.951 (19.84) | 0.977 (16.81)
  Tumor Necrosis Factor, Week 4, n=9, 27: number analyzed (Participants) | 9 | 27
  Tumor Necrosis Factor, Week 4, n=9, 27 | 0.933 (17.70) | 0.871 (48.19)
  Tumor Necrosis Factor, Week 6, n=7, 27: number analyzed (Participants) | 7 | 27
  Tumor Necrosis Factor, Week 6, n=7, 27 | 1.087 (36.81) | 0.929 (21.48)
  Tumor Necrosis Factor, Week 8, n=7, 25: number analyzed (Participants) | 7 | 25
  Tumor Necrosis Factor, Week 8, n=7, 25 | 1.110 (25.33) | 0.930 (20.85)
  Tumor Necrosis Factor, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Tumor Necrosis Factor, Week 12, n=7, 24 | 1.021 (38.53) | 0.969 (29.74)
  Tumor Necrosis Factor,12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Tumor Necrosis Factor,12-Week FU, n=7, 21 | 1.619 (180.16) | 1.057 (34.72)

18. Primary Outcome: Change From Baseline in Safety Biomarkers: 3B-Cholestenoic Acid, Surfactant Protein D
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Safety biomarkers included analysis of 3B-Cholestenoic Acid and Surfactant Protein D. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Week 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of safety biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of safety biomarker
  3B-Cholestenoic Acid, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  3B-Cholestenoic Acid, Week 12, n=7, 24 | 1.012 (16.52) | 1.094 (19.45)
  3B-Cholestenoic Acid, Week 22, n=7, 22: number analyzed (Participants) | 7 | 22
  3B-Cholestenoic Acid, Week 22, n=7, 22 | 1.020 (20.25) | 1.009 (22.67)
  Surfactant Protein D, Week 12, n=7, 24: number analyzed (Participants) | 7 | 24
  Surfactant Protein D, Week 12, n=7, 24 | 1.003 (23.10) | 1.134 (27.96)
  Surfactant Protein D, 12-Week FU, n=7, 21: number analyzed (Participants) | 7 | 21
  Surfactant Protein D, 12-Week FU, n=7, 21 | 1.140 (45.71) | 0.985 (31.32)

19. Primary Outcome: Change From Baseline in Safety Biomarkers: KL-6 Antigen
Description: Blood samples were collected and analyzed for markers which may be predictive of rheumatoid arthritis disease activity. Safety biomarker included analysis of KL-6 Antigen. Baseline was defined at Day 1. Change from Baseline was calculated as ratio of Baseline value to post-dose value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Week 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of safety biomarker
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Ratio of safety biomarker
  Week 12, n=6, 24: number analyzed (Participants) | 6 | 24
  Week 12, n=6, 24 | 1.416 (220.58) | 1.099 (66.17)
  12-Week FU, n=6, 21: number analyzed (Participants) | 6 | 21
  12-Week FU, n=6, 21 | 0.937 (62.43) | 1.024 (93.56)

20. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect and associated with liver injury and impaired liver function. An AESI include serious infections, opportunistic infections, neutropenia, respiratory events, pulmonary alveolar proteinosis, hypersensitivity reactions, injection site reactions, persistent cough or dyspnea.
Time Frame: Up to 12-Week FU (Week 22)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Participants
  Any AEs | 4 | 11
  Any SAEs | 0 | 0
  AESI | 0 | 1

21. Secondary Outcome: Number of Participants Who Tested Positive for Anti-GSK3196165 Binding Antibody Detection at Any Time Post-Baseline
Description: Immunogenicity samples for determination of anti-drug-antibody (ADA) were collected. The presence of treatment emergent ADA was determined using a GSK3196165 bridging style ADA assay with a bio-analytically determined cut point determined during assay validation. Samples taken after dosing with GSK3196165 that had a value at or above the cut-point was considered potentially treatment-emergent ADA-positive. The immunogenicity population consisted of all participants in the ITT population, who had at least one valid immunogenicity assessment.
Time Frame: Up to 12-Week FU (Week 22)
Population: Immunogenicity Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Participants | 0 | 0

22. Secondary Outcome: Change From Baseline in Synovitis as Assessed by Outcome Measures in Rheumatology (OMERACT) Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) in the Most Affected Hand/Wrist
Description: For synovitis a total of 8 joints were evaluated. Individual joint scores range from 0-3, where 0= normal, 1=mild, 2=moderate and 3=severe. The final synovitis score is the sum of the individual joint scores. Total score range from 0 (best) to 24 (worst). If an individual location is scored either 'Not Visible' or 'Surgically Modified' then the score for that location was set to missing. Missing joint scores was imputed as the mean of the non-missing joint scores. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Repeated measures analysis adjusted for synovitis score baseline value, treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Data has been presented for Median and 95% credible interval. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Scores on a scale
  Week 4, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 4, n=6, 12 | 0.05 [-1.92 to 1.95] | -0.07 [-1.19 to 1.12]
  Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  Week 12, n=5, 21 | 0.84 [-1.57 to 3.12] | -1.33 [-2.54 to -0.13]
  12-Week FU, n=7, 19: number analyzed (Participants) | 7 | 19
  12-Week FU, n=7, 19 | 1.13 [-1.32 to 3.55] | -1.13 [-2.47 to 0.20]
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Week 4, For Posterior Probability Difference <0; Test type: Other; p = 0.547, Repeated Measures Bayesian Model; Median Difference (Net) = -0.13, 95% CI 2-sided [-2.32 to 2.23]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Week 12, For Posterior Probability Difference <0; Test type: Other; p = 0.948, Repeated Measures Bayesian Model; Median Difference (Net) = -2.18, 95% CI 2-sided [-4.77 to 0.51]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU, For Posterior Probability Difference <0; Test type: Other; p = 0.949, Repeated Measures Bayesian Model; Median Difference (Net) = -2.28, 95% CI 2-sided [-5.02 to 0.45]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 180 mg; Week 4, For Posterior Probability Difference >0; Test type: Other; p = 0.453, Repeated Measures Bayesian Model; Median Difference (Net) = -0.13, 95% CI 2-sided [-2.32 to 2.23]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; Week 12, For Posterior Probability Difference >0; Test type: Other; p = 0.052, Repeated Measures Bayesian Model; Median Difference (Net) = -2.18, 95% CI 2-sided [-4.77 to 0.51]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU, For Posterior Probability Difference >0; Test type: Other; p = 0.051, Repeated Measures Bayesian Model; Median Difference (Net) = -2.28, 95% CI 2-sided [-5.02 to 0.45]

23. Secondary Outcome: Change From Baseline in Osteitis as Assessed by OMERACT RAMRI Scoring System in the Most Affected Hand/Wrist
Description: For bone edema/osteitis a total of 25 locations was evaluated. Individual location scores ranged from 0-3, where, 0: no edema; 1: 1-33% of bone edematous; 2: 34-66% of bone edematous; 3: 67-100% of bone edematous. Final bone edema/osteitis score is sum of individual location scores. Total score ranged from 0 (best) to 75 (worst). Baseline was defined at Day 1. Change from Baseline was calculated by subtracting post-dose value from Baseline value. If an individual location was scored either 'Not Visible' or 'Surgically Modified' or 'Not Assessable' then the score for that location was set to be missing. Missing joint scores was imputed as mean of non-missing location scores. Repeated measures analysis adjusted for Bone Edema/Osteitis Score baseline value, treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Scores on a scale
  Week 4, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 4, n=6, 12 | -0.1 (0.11) | -0.1 (0.06)
  Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  Week 12, n=5, 21 | 0.0 (1.04) | -0.8 (0.56)
  12-Week FU, n=7,19: number analyzed (Participants) | 7 | 19
  12-Week FU, n=7,19 | 0.5 (1.33) | -0.9 (0.74)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Week 4; Test type: Other; p = 0.940, Repeated measures analysis; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Week 12; Test type: Other; p = 0.521, Repeated measures analysis; Mean Difference (Net) = -0.8, 95% CI 2-sided [-3.2 to 1.6]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU; Test type: Other; p = 0.396, Repeated measures analysis; Mean Difference (Net) = -1.3, 95% CI 2-sided [-4.4 to 1.8]

24. Secondary Outcome: Change From Baseline in Erosion as Assessed by OMERACT RAMRI Scoring System in the Most Affected Hand/Wrist
Description: For bone erosion a total of 25 locations were evaluated. Individual location scores range from 0-10, where, 0: no erosion; 1: 1-10% of bone eroded and 10: 91-100% of bone eroded. The final bone erosion score is the sum of the individual location scores. The total score ranged from 0 (best) to 250 (worst). If an individual location was scored either 'Not Visible' or 'Surgically Modified' or 'Not Assessable' then the score for that location was set to be missing. Missing joint scores was imputed as the mean of the non-missing location scores. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Analysis was performed using repeated measures analysis adjusted for Bone Erosion Score baseline value, treatment group, disease duration (<=2 or >2 years), visit and treatment group. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles.
Time Frame: Baseline and Weeks 4, 12, 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Scores on a scale
  Week 4, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 4, n=6, 12 | 0.2 (0.49) | 0.3 (0.30)
  Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  Week 12, n=5, 21 | 0.8 (0.50) | 0.4 (0.26)
  12-Week FU, n=7, 19: number analyzed (Participants) | 7 | 19
  12-Week FU, n=7, 19 | 1.5 (0.47) | 0.5 (0.27)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Week 4; Test type: Other; p = 0.945, Repeated measures analysis; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.1 to 1.2]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Week 12; Test type: Other; p = 0.475, Repeated measures analysis; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.5 to 0.7]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU; Test type: Other; p = 0.086, Repeated measures analysis; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.0 to 0.1]

25. Secondary Outcome: Change From Baseline in Synovitis as Assessed by Rheumatoid Arthritis MRI Quantitative (RAMRIQ) Assessment in the Most Affected Hand/Wrist
Description: RAMRIQ is an automated volume quantification assessment. RAMRIQ assessed same pathologies and joints (except metacarpophalangeal joint [MCP1]) as RAMRIS allowing for direct comparison of results obtained using the two methods. Bones were automatically identified in pre-contrast, coronal T1 images using active appearance modelling (AAMs). Joint capsules and soft tissues were also segmented with AAMs, providing consistent 3D regions of interest (ROI) for synovial enhancement across all time points. Synovial volume was calculated as voxels that enhance within each ROI. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Repeated measures analysis adjusted for Synovitis baseline value, treatment group, disease duration (<=2 or >2 years), visit and treatment group by visit interaction. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 4, 12 and 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Milliliters
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Milliliters
  Week 4, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 4, n=6, 12 | 34.1 (1052.52) | 245.5 (776.24)
  Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  Week 12, n=5, 21 | -912.3 (1405.77) | -1417.0 (671.54)
  12-Week FU, n=7, 19: number analyzed (Participants) | 7 | 19
  12-Week FU, n=7, 19 | 364.0 (1372.20) | -1172.1 (844.13)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Week 4; Test type: Other; p = 0.874, Repeated measures analysis; Mean Difference (Net) = 211.4, 95% CI 2-sided [-2589.2 to 3012.0]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Week 12; Test type: Other; p = 0.749, Repeated measures analysis; Mean Difference (Net) = -504.8, 95% CI 2-sided [-3730.4 to 2720.9]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU; Test type: Other; p = 0.352, Repeated measures analysis; Mean Difference (Net) = -1536.0, 95% CI 2-sided [-4884.2 to 1812.1]

26. Secondary Outcome: Change From Baseline in Osteitis as Assessed by RAMRIQ Assessment in the Most Affected Hand/Wrist
Description: RAMRIQ is an automated volume quantification assessment for edema volume. RAMRIQ assessed the same pathologies and joints (except MCP1) as RAMRIS, allowing for direct comparison of results obtained using the two methods. Bones were automatically identified in pre-contrast, coronal T1 images using AAMs. Joint capsules and soft tissues were also segmented with AAMs, providing consistent 3D ROI for synovial enhancement across all time points. Edema volume was defined as non-erosion contrast-enhancing voxels inside the bone. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 4, 12 and 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Milliliters
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Milliliters
  Week 4, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 4, n=6, 12 | -0.0045 (0.0102) | 0.0084 (0.0057)
  Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  Week 12, n=5, 21 | -0.0045 (0.0035) | -0.0009 (0.0019)
  12-Week FU, n=7, 19: number analyzed (Participants) | 7 | 19
  12-Week FU, n=7, 19 | -0.0038 (0.0016) | -0.0027 (0.0009)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Week 4; Test type: Other; p = 0.291, Repeated measures analysis; Mean Difference (Net) = 0.0128, 95% CI 2-sided [-0.0123 to 0.0380]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Week 12; Test type: Other; p = 0.375, Repeated measures analysis; Mean Difference (Net) = 0.0036, 95% CI 2-sided [-0.0046 to 0.0118]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU; Test type: Other; p = 0.588, Repeated measures analysis; Mean Difference (Net) = 0.0010, 95% CI 2-sided [-0.0028 to 0.0049]

27. Secondary Outcome: Change From Baseline in Erosion as Assessed by RAMRIQ Assessment in the Most Affected Hand/Wrist
Description: RAMRIQ is an automated volume quantification assessment for erosion volume. RAMRIQ assessed the same pathologies and joints (except MCP1) as RAMRIS, allowing for direct comparison of results obtained using the two methods. Bones were automatically identified in pre-contrast, coronal T1 images using AAMs. Joint capsules and soft tissues were also segmented with AAMs, providing consistent 3D ROI for synovial enhancement across all time points. Erosion volume was identified inside the bone surfaces using voxel-based classification. The volume of BME and erosions was normalised to total bone volume for statistical analysis. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-dose value from the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Weeks 4, 12 and 12-Week FU (Week 22)
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Milliliters
Arm/Group | Placebo | GSK3196165 180 mg
Number analyzed (Participants) | 11 | 28
Milliliters
  Week 4, n=6, 12: number analyzed (Participants) | 6 | 12
  Week 4, n=6, 12 | 0.0007 (0.0012) | 0.0006 (0.0008)
  Week 12, n=5, 21: number analyzed (Participants) | 5 | 21
  Week 12, n=5, 21 | 0.0003 (0.0011) | -0.0000 (0.0006)
  12-Week FU, n=7, 19: number analyzed (Participants) | 7 | 19
  12-Week FU, n=7, 19 | -0.0002 (0.0023) | 0.0003 (0.0013)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 180 mg; Week 4; Test type: Other; p = 0.915, Repeated measures analysis; Mean Difference (Net) = -0.0002, 95% CI 2-sided [-0.0033 to 0.0029]
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 180 mg; Week 12; Test type: Other; p = 0.771, Repeated measures analysis; Mean Difference (Net) = -0.0004, 95% CI 2-sided [-0.0028 to 0.0021]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; 12-Week FU; Test type: Other; p = 0.850, Repeated measures analysis; Mean Difference (Net) = 0.0005, 95% CI 2-sided [-0.0048 to 0.0058]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from start of study treatment up to 12-Week FU (Week 22).
Description: ITT Population was used for the analysis of safety data.
Arm/Group | Placebo | GSK3196165 180 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/28
Other Adverse Events (participants affected / at risk) | 4/11 | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | GSK3196165 180 mg (N=28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Weight increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02799472/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT02799472/SAP_001.pdf